

#### 2015-0013-00US1

A MULTI-CENTER, OPEN-LABEL, PHASE 1/1B CLINICAL STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND ANTICANCER ACTIVITY OF FRUQUINTINIB IN PATIENTS WITH ADVANCED SOLID TUMORS

| <b>Author:</b> | | | |
|----------------|------------|--------------------|-----------|
| <b>Version</b> | Number and | <b>Date:</b> V2.5, | 18FEB2022 |

 Document:
 Version Number:
 2.5

 Author:
 Version Date:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005



## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V2.5 (Dated 18Feb2021) for Protocol 2015-013-00US1.

| | Name | Signature | Date (DDMMYYYY) |
|-----------|-------|-------------|---------------------------------|
| Author: | | e-signature | Please refer to log on Wingspan |
| Position: | | | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMMYYYY) |
|--------------|-------------------|-----------|-----------------|
| Approved By: | | Signature | Date (DDMMYYYY) |
| Position: | | | |
| Company: | Hutchison Medi Ph | arma Ltd. | |
| Approved By: | | Signature | Date (DDMMYYYY) |
| Position: | | | |
| Company: | Hutchison Medi Ph | arma Ltd. | |

| Document: | | |
|---------------------------|------------------------|-----------|
| Author: | Version Number: | 2.5 |
| | Version Date: | 18Feb2022 |
| Template No.: | Reference: CS_WI_BS005 | |
| Effective Date: 02Dec2019 | | |


## **OUTPUT TEMPLATES SIGNATURE PAGE**

Output Templates V2.5 (Dated 18Feb2022) for Protocol 2015-013-00US1.

| | Name | Signature | Date (DDMMYYYY) |
|-----------|-------|-------------|---------------------------------|
| Author: | | e-signature | Please refer to log on Wingspan |
| Position: | | | - |
| Company: | IQVIA | _ | |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMMYYYY) |
|--------------|-------------|-----------------|-----------------|
| Approved By: | | Signature | Date (DDMMYYYY) |
| Position: | | | |
| Company: | Hutchison M | edi Pharma Ltd. | |
| Approved By: | | Signature | Date (DDMMYYYY) |
| Position: | | | |
| Company: | Hutchison M | edi Pharma Ltd. | |

| Document: | |
|---------------------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |
| Effective Date: 02Dec2019 | |



## **MODIFICATION HISTORY**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| 0.1 | 10Jan2018 | | Not Applicable – First Version |
| 0.2 | 15Mar2018 | | Revise 3.1 section according to protocol version 2 Revise the REAS according to protocol version 2 Add the FAS according to the requirement for analysis Delete the shift table for low, high, normal according to protocol |
| 0.3 | 24Jan2019 | | Add the definition of OS and PFS at 12 weeks Revise the population set of REAS to EAS. Add the definition of subsequent anticancer therapy. Delete the shift from baseline analysis of ECOG PS. Global changes according to protocol version 3. |
| 1.0 | 30Jan2019 | | Upgrade version, no updates. |
| 1.0 | 17Jan2020 | | Updating SAP & Shell according to sponsor' comments |
| 1.1 | 11Feb2020 | | Updating SAP & Shell according to sponsor' comments |
| | 03Mar2020 | | Update Table 14.1.1.1, Table 14.1.6.1, source listing of Table 14.1.6.2, |
| | 09Mar2020 | | Update shell of "Listing 16.2.7.2" |
| | 12Mar2020 | | Revise source listing of Table 14.1.3, update section 7.3 |
| | 16Mar2020 | | Update notes to programmer of Listing 16.2.7.3 Update layout of Listing 16.2.1.1, 16.2.1.2 and 16.2.6.5 |
| | 17Mar2020 | | Updating Source of Table 14.1.2 and notes to programmer of Listing 16.2.9.1.1 |

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005



| | 07Apr2020 | - Updating Listing 16.2.1.2, 16.2.3.1, |
|-----|------------|---------------------------------------------|
| | 07Apr2020 | 16.2.4.2, 16.2.5.1.1, 16.2.5.2, 16.2.5.1.3, |
| | | 16.2.5.6, 16.2.7.2, 16.2.6.4, 16.2.7.7; |
| | | Table 14.1.4.3.2, 14.3.1.2, 14.3.1.3.2 |
| | | - Updating footnote of Listing 16.2.4.2, |
| | | 16.2.5.1.2, 16.2.5.2, 16.2.5.3; Table |
| | | 14.3.1.6.2, 14.3.1.7.3, 14.3.1.8.3, |
| | | - Updating note to programmer of Table |
| | | 14.3.1.11.3, 14.3.1.12.3, |
| | | - Typo: Listing 16.2.4.2, 16.2.5.1.2, |
| | | - Revision of table caption: 14.2.1.1, |
| | | 14.2.2.1, 14.2.3.1, 14.2.4.1, 14.2.5.1 |
| | | - Adding Table 14.2.1.2, 14.2.2.2, |
| | | 14.2.3.2, 14.2.4.2, 14.2.5.2, 14.4.1, |
| | | 14.4.2 |
| | | - Adding Figure 14.2.1.2, 14.2.2.2, |
| | | 14.2.3.2, 14.2.4.2, and 14.4.1 |
| | | - SAP update: 18.2.1 |
| 1.2 | 15Oct2020 | - Revision done for amended protocol |
| 1.2 | 130012020 | V.4.0 |
| | | -Wording change on replacing 'subject' |
| | | with 'patient' |
| | | -Typos |
| | | -Output Conventions |
| | | -Revisions were done in almost all |
| | | sections except for section 4.2, 6, 7.1, |
| | | 7.2, 7.3.3-7.5, 8, and 14. |
| 2.0 | 23Nov2020 | Revision according to sponsor's |
| | | comments |
| | 30Nov2020 | - Revisions of format and typos |
| | | - Remove one blank page |
| | 04Dec2020 | - Remove section 2.3 to Appendix 1 |
| | | - Re-number all appendices |
| | | - Revisions of section 3, 5.7, 6.2, 6.3.1, |
| | | 6.3.2, 7-12, 13.2, 14, 15.1, 16.1.5, 16.2 |
| | | - Changes on wording according to |
| | | sponsor's comments |
| | 08Dec2020 | Revise SI unit of: Alkaline Phosphatase, |
| | | Aspartate Aminotransferase, Alanine |
| | | Aminotransferase |
| | 09Dec2020 | Update Appendix 4 |
| | 10Dec2020 | Update section 2.4 and 17.4.4 |
| | 1010002020 | Opuate section 2.7 and 17.4.4 |

Document:

Author:

Version Number: 2.5


Template No.: Reference: CS\_WI\_BS005


| | 16Dec2020 | <ul> <li>Section 17.7 and corresponding shell</li> <li>Update some inconsistencies based on shell</li> <li>Specify cut-off date on header</li> <li>Separate Table 14.1.1.1 into 2 tables and update footnote separately</li> <li>Footnote update for some tables</li> <li>Update Appendix 4</li> <li>typo correction</li> </ul> |
|---|---|---|
| | 18Dec2020 | Date update |
| 2.2 | 02Jul2021 | Update Appendix 2: Presentation of Treatment Groups |
| 2.3 | 16Nov2021 | Date update |
| 2.4 | 13Dec2021 | <ul> <li>Version and date updated</li> <li>Updated format of Appendix 4, 5 and 6</li> <li>Updated table 2 and AESI description in section 17.2.6</li> <li>Removed additional blank</li> <li>Updated listing 16.2.9.6</li> <li>Pharmacokinetic Blood Sample (Pharmacokinetic Analysis Set) to listing 16.2.9.6 COVID-19 Visit Impact (Safety Analysis Set)</li> </ul> |
| 2.5 | 18Feb2022 | <ul> <li>Version and date updated</li> <li>Update the AESI list of table in</li> <li>Appendix 5, the old list is the MedDRA</li> <li>24.0, and the updated list is using</li> <li>MedDRA 24.1.</li> </ul> |

Document: Author: Version Number: 2.5 Version Date: 18Feb2022 Template No.: Reference: CS\_WI\_BS005





#### **TABLE OF CONTENTS**

| Statisti | tical Analysis Plan Signature Page | 2 |
|----------------|------------------------------------|-----|
| Outpu | ıt Templates Signature Page | 3 |
| MOD | DIFICATION HISTORY | 4 |
| Table ( | of Contents | 7 |
| LIST | OF ABBREVIATIONS | 10 |
| 1. | Introduction | 12 |
| 1.1. | | |
| 1.1.1 | 1. Dose Escalation Phase | 12 |
| 1.1.2 | 2. Dose Expansion Phase | 12 |
| 1.2. | Secondary Objectives | 12 |
| 1.2.1 | 1. Dose Escalation Phase | 12 |
| 1.2.2 | 2. Dose expansion Phase | 12 |
| 2. | Study Design | 13 |
| 2.1. | | |
| 2.2. | | |
| 2.3. | 1 | |
| 2.3.1 | $\mathcal{J}$ | |
| 2.3.2 | | |
| 2.4. | | |
| 3. | Dlamad Analysis | 16 |
| <b>3.</b> 3.1. | Planned Analyses Interim Analysis | |
| 3.1. | | |
| 3.2. | 1 mai 7 mai y sis | 1 / |
| 4. | Analysis Sets | |
| 4.1. | L J | |
| 4.2. | | |
| 4.3. | $\mathcal{E}$ | |
| 4.4. | Efficacy Analysis Set [EAS] | 17 |
| 5. | General Considerations | 18 |
| 5.1. | | |
| 5.2. | | |
| 5.3. | | |
| 5.4. | | |
| 5.5. | e | |
| 5.6. | | |
| 5.7. | Software Version | 19 |
| 6. | Statistical Considerations | 19 |
| Docum | nent: | |

Author:


Reference: CS\_WI\_BS005

2.5


18Feb2022

Effective Date: 02Dec2019

Template No.:



| 6.1. | Adjustments for Covariates and Factors to be Inc | cluded in Analyses | 19 |
|---|---|---|---|
| 6.2. | Multicenter Studies | | |
| 6.3. | Missing data | | |
| 6.3.1. | Missing Dates Information of Study Treatment. | | |
| 6.3.2. | Missing or Incomplete Date Information for Adv | verse Event Date | 20 |
| 6.3.3. | Missing or Incomplete Date Information for con | comitant Medication/ Procedure | 22 |
| 6.3.4. | Missing or Incomplete Date Information for Prin 22 | mary Diagnosis Date and Metastatic D | iagnosis Date |
| 6.3.5. | Missing or Incomplete Date Information for Effi | icacy Data | 22 |
| 6.4. | Multiple Comparisons/ Multiplicity | | |
| 6.5. | Examination of Subgroups | | 22 |
| 7. Ou | put Presentations | | 23 |
| | position and Withdrawals | | |
| 8.1. | Enrollment | | |
| 8.2. | Patient status at treatment and study completion | | 24 |
| 9. Pro | tocol Deviation | | 24 |
| 10. Der | nographic and other Baseline Characteristics Derivations | | |
| 11. Sur | gical and Medical History | | 25 |
| | cology History | | |
| 12.1. | Derivations | | 26 |
| 13. On | cological Therapies | | 26 |
| 13.1. | Prior oncological therapy | | 26 |
| 13.2. | Subsequent Oncology Therapy | | 27 |
| 14. Me | dications and Procedures | | 27 |
| 14.1. | Prior and Concomitant Medication | | |
| 14.2. | Concomitant procedures | | 28 |
| 15. Stu | dy Medication Exposure | | 28 |
| 15.1. | Exposure to study medication | | |
| 15.2. | Study Medication Compliance | | 29 |
| 15.3. | Derivations | | 29 |
| | cacy Outcomes | | |
| 16.1. | Primary Efficacy Variable(s) & Derivation(s) | | |
| 16.1.1. | Best Overall Response (BOR) | | |
| 16.1.2. | Objective Response Rate (ORR) | | |
| 16.1.3. | Duration of Response (DoR) | | |
| 16.1.4.<br>16.1.5. | Duration Control Rate (DCR)<br>Progression Free Survival (PFS) | | |
| 16.1.5. | Overall Survival (OS) | | |
| 16.1.6. | Tumor Shrinkage | | |
| 16.1.7. | Analysis of Efficacy Variable(s) | | |
| Document: | | | |
| Author | | Version Number: | 2.5 |
| Author: | | Version Number: Version Date: | 2.5<br>18Feb2022 |
| Template N | 0. | Reference: CS_WI_BS005 | 101 602022 |
| · ciribiate I | · · · | 1 (CICICITOC. OC_VVI_DOUD) | |



| 17. Safe | ty Outcomes | .34 |
|---|---|---|
| 17.1. | DLTs | .34 |
| 17.2. | Adverse Events | .35 |
| 17.2.1. | All TEAEs | |
| 17.2.2. | TEAEs Leading to Dose Interruption or Reduction | .36 |
| 17.2.3. | TEAEs Leading to Discontinuation of Study Drug | .36 |
| 17.2.4. | Serious Adverse Events | |
| 17.2.5. | Adverse Events Leading to Death | |
| 17.2.6. | Adverse Events Of Special Interest (AESI) | |
| 17.3. | Deaths | |
| 17.4. | Laboratory Evaluations | .37 |
| 17.4.1. | Laboratory Specific Derivations | |
| 17.4.2. | CTCAE Grading for Laboratory Data | |
| 17.4.3. | Laboratory Reference Ranges | .39 |
| 17.4.4. | Potential Drug-Induced Liver Injury (DILI) | .39 |
| 17.5. | ECG Evaluations | |
| 17.5.1. | ECG Specific Derivations. | |
| 17.5.2. | Markedly Abnormal Criteria | |
| 17.6. | Vital Signs | |
| 17.6.1. | Vital Signs Specific Derivations | |
| 17.6.2. | Vital Signs Markedly Abnormal Criteria | |
| 17.7. | Physical Examination | .43 |
| 17.8. | Other Safety Assessments | |
| 17.8.1. | ECOG Performance Status | .43 |
| 17.8.2. | Echocardiogram | .43 |
| 17.8.3. | Pregnancy Test | .43 |
| 17.8.4. | Tumor Marker | .43 |
| 17.8.5. | Impact of COVID-19 | .44 |
| 18. Refe | erences | .44 |
| APPENDIX | X 1. Schedule of Events | .45 |
| A DDENIDI | VA Durance Comment of | 47 |
| APPENDIZ | X 2. Programming Conventions for Outputs | .4/ |
| APPENDIX | X 3. Best Overall Response When Confirmation of CR and PR are Required | 49 |
| APPENDIX | K 4. Visit-Window Mapping | .51 |
| APPENDIX | X 5. MedDRA (Version 24.1) Preferred Term List for AESI Categories | .54 |
| A PPENDI | X 6. Clinical Laboratory Parameters CTCAE Criteria | 72 |

Document:

Author:


2.5


18Feb2022

Template No.: Effective Date: 02Dec2019

Reference: CS\_WI\_BS005



 Statistical Analysis Plan

## **LIST OF ABBREVIATIONS**

| Terms and | |
|---------------|-------------------------------------------------------------|
| Abbreviations | Definition |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| ALT | Alanine Aminotransferase/Glutamic-Pyruvic Transaminase |
| APTT | Activated Partial Thromboplastin time |
| AST | Aspartate Aminotransferase/Glutamic-Oxalacetic Transaminase |
| ATC | Anatomical Therapeutic Classification |
| BC | Breast Cancer |
| BMI | Body Mass Index |
| BOR | Best Overall Response |
| CEA | Carcino-Embryonic Antigen |
| CR | Complete Response |
| CS | Clinically Significant |
| CTCAE | Common Terminology Criteria for Adverse Event |
| CTMS | Clinical Trial Management System |
| DCR | Disease Control Rate |
| DLT | Dose-Limiting Toxicity |
| DoR | Duration of Response |
| DILI | Drug Induced Liver Injury |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram |
| ECOG PS | Eastern Cooperative Oncology Group Performance Status |
| eCRF | Electronic Case Report Form |
| ENR | All Patients Enrolled Set |
| HR | Hormone Receptor |
| INR | International Normalized Ratio |
| LLQ | Lower Limit of Quantification |
| mCRC | Metastatic Colorectal Cancer |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MUGA | Multi-Gated Acquisition |
| NCI | National Cancer Institute |

Document:


Template No.: Reference: CS\_WI\_BS005




NCS Not Clinically Significant

NE Not Evaluable

NSCLC Non-Small Cell Lung Cancer
ORR Objective Response Rate

OS Overall Survival
PD Progressive Disease

PFS Progressive Free Survival
PID Percentage Intended Dose

PLT Blood platelet count

PR2D Recommended Phase 2 Dose

PR Partial Response
RD Relative Dose
PT Preferred Term

QD Quaque Die/ Once Daily RDI Relative Dose Intensity

RECIST Response Evaluation Criteria in Solid Tumors

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Safety Analysis Set

SD Stable Disease

SMQ Standardized MedDRA Queries

SOC System Organ Class STD Standard Deviation

TEAE Treatment-Emergent Adverse Event

TEAESI Treatment-Emergent Adverse Event of Special Interest

TNBC Triple-Negative Breast Cancer
TSH Thyroid stimulating hormone

ULN Upper Limit of Normal

ULQ Upper Limit of Quantification

VEGF Vascular Endothelial Growth Factor

WHO DDE World Health Organization Drug Dictionary Enhanced

Document:


Template No.: Reference: CS\_WI\_BS005

#### 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of efficacy and safety data for Protocol 2015-013-00US1. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol Version 4.0 (Amendment 4), dated 09 Jan 2020. The Pharmacokinetics (PK) and pharmacodynamics analyses will not be performed by IQVIA Biostatistics (BIOS) and therefore are not documented in this SAP.

#### 1.1. PRIMARY OBJECTIVE

#### 1.1.1. DOSE ESCALATION PHASE

The primary objective of the dose escalation phase is to evaluate the safety and tolerability of fruquintinib in patients with advanced solid tumors and to determine the recommended Phase 2 dose (RP2D).

#### 1.1.2. DOSE EXPANSION PHASE

The primary objective of the dose expansion phase is to evaluate the anticancer activity of fruquintinib at the recommended RP2D from the dose escalation phase, in patients with advanced solid tumors.

#### 1.2. SECONDARY OBJECTIVES

#### 1.2.1. DOSE ESCALATION PHASE

The secondary objectives of the dose escalation phase are:

- To evaluate the PK characteristics of multiple dose fruquintinib and to investigate the metabolite profile of fruquintinib in the plasma of patients with solid tumors (The detailed analysis method will not be documented in this document).
- To evaluate anticancer activity of fruquintinib in patients with solid tumors according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (Eisenhauer et al., 2009).

#### 1.2.2. DOSE EXPANSION PHASE

The secondary objectives of the dose expansion phase are:

- To evaluate anticancer efficacy of fruquintinib, as assessed by Objective response rate (ORR), disease control rate (DCR), duration of response (DoR), progression free survival (PFS) and overall survival (OS).
- To evaluate the PK characteristics of multiple dose fruquintinib and to investigate the metabolite profile of fruquintinib in plasma.
- To evaluate the safety of fruquintinib.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

 Effective Date:
 02Dec2019



#### 2. STUDY DESIGN

The study is an open-label phase 1/1b study of fruquintinib comprised of a dose escalation phase that will enroll patients with advanced solid tumors of any type, and a dose expansion phase that will enroll patients with advanced solid tumors of any type (Cohort A) and in patients with refractory metastatic colorectal cancer (mCRC, Cohort B and C), or breast cancer (BC, Cohort D and E) (see study schema below).



Approximately 128 patients will be enrolled in this dose escalation/dose expansion study. Approximately 12 patients will be enrolled in the dose escalation phase, and approximately 116 additional patients (6 with advanced solid tumors of any type and 40 with refractory mCRC who progressed on TAS-102 and/or regorafenib, 40 with mCRC who had not received TAS-102 or regorafenib, 15 with refractory HR+/HER2- mBC, and 15 with advanced, refractory triple-negative breast cancer (TNBC) will be enrolled in the dose expansion phase.

#### 2.1. DOSE ESCALATION PHASE

Approximately 12 evaluable patients will be enrolled. The actual number of patients will depend on the occurrence of dose-limiting toxicities (DLTs) as well as the Maximum Toxicity Dose (MTD) level reached in this trial. MTD is the highest dose at which no more than 1 of the 6 patients in each cohort of the dose escalation phase develops a DLT. If 2 or more of 6 patients in each cohort of the dose escalation phase develop DLT at a particular dose level, that dose has exceeded the MTD. The dose levels to be investigated are 3 mg and 5 mg once daily (QD), 3 weeks on/1 week off.




The definition of DLTs and the DLT assessment window is provided in <u>section 17.1</u> and the definition of a DLT evaluable patient is provided in <u>section 4.3</u>.

To investigate DLT, 6 DLT-evaluable patients will be firstly enrolled in the phase and will be treated with fruquintinib 3 mg QD (3 weeks on/1 week off) orally. If no more than 1 DLT occurs during the DLT observational window (i.e. from Day 1 – 28 in Cycle 1) among the 6 patients, the trial will continue to enroll another 6 patients in the next dose cohort in which fruquintinib 5 mg QD (3 weeks on / 1 week off) will be tested. Safety monitoring and evaluation for the dose escalation phase will be carried out by the Safety Review Committee (SRC). If no more than 1 patient at the dose level of 5 mg QD experiences a DLT, the dose escalation phase is completed, and the expansion phase of the study will be conducted. Upon the completion of the dose escalation phase, the SRC will review aggregated safety and PK data and then select a fruquintinib dose as the RP2D for the expansion phase of the trial. Prior to confirmation of a DLT, if a patient has received any prophylactic medical intervention or missed 4 or more fruquintinib dose during the DLT observational window, the patient is not DLT evaluable and will be replaced. If a patient does not meet the definition of DLT evaluable patient criterion during the DLT observation period, the patient will be replaced. Patients who have completed the DLT observation period (Days 1 – 28, Cycle 1) and are deemed to be benefiting from the fruquintinib treatment at the investigator's discretion may continue the fruquintinib treatment until disease progression, death, intolerable toxicity, or at investigator's discretion that the patient can no longer benefit from the study drug.

Patients will be followed until death or study completion, which is defined as the CRF form "End of Study" is filled.

#### 2.2. DOSE EXPANSION PHASE

Once the RP2D is determined, patients may enroll into one of the following cohorts and will receive fruquintinib at the RP2D.

- Cohort A: Patients with advanced, refractory solid tumors of any type.
- Cohort B: Patients with refractory mCRC who have progressed on all standard chemotherapies and relevant biologics and have also progressed on, or had intolerable toxicity with, at least 1 FDA-approved third-line therapy (TAS-102 or regorafenib).
- Cohort C: Patients with refractory mCRC who have progressed on all standard chemotherapies and relevant biologics and have not received prior TAS-102 or regorafenib.
- Cohort D: Patients with hormone-receptor positive (ER+ and/or PR+)/Her2-metastatic breast cancer who have progressed on at least two line of prior systemic therapy.
- Cohort E: Patients with advanced TNBC who have progressed on at least one cytotoxic therapy in the metastatic setting

Document:

Author:


18Feb2022

Template No.:

Reference: CS\_WI\_BS005

Effective Date: 02Dec2019


The safety of all enrolled patients will be closely monitored from the first day of fruguintinib dosing until 30 days after the last dose. All serious adverse events (SAEs) should be reported from the day the informed consent form (ICF) is signed through 30 days after last dose regardless of relationship to study drug. All AEs will be graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V4.03.

In the dose expansion phase, tumor response will be assessed according to RECIST Version 1.1 (Eisenhauer et al., 2009) at screening, and at study visits according the Schedule of Events (Appendix A in the protocol). Confirmation of complete response (CR) and partial response (PR) is required at no less than 4-week intervals between the date of initial response and the confirmation assessment date.

Patients will be followed until death or study completion.

#### 2.3. STUDY ENDPOINTS

#### 2.3.1. DOSE ESCALATION PHASE

- Primary Endpoints: The primary endpoint of the dose escalation phase is the incidence of DLT in each cohort.
- Secondary endpoints: The objective response rate (ORR), disease control rate (DCR), duration of response (DoR), and progression free survival (PFS) according to RECIST Version 1.1 (Eisenhauer et al., 2009), overall survival (OS) and percentage change from baseline in tumor size.

#### 2.3.2. DOSE EXPANSION PHASE

- Primary endpoint: PFS
- Secondary endpoints:
  - Efficacy analysis: ORR, DCR, DoR, PFS according to RECIST Version 1.1 (Eisenhauer et al., 2009), OS and percentage change in tumor size from baseline.
  - Safety analysis: the incidence and severity of adverse events (AEs), physical examinations, vital signs, laboratory test results, 12-lead electrocardiogram, and echocardiogram.

Document:

Author: Version Number:

18Feb2022

2.5

Reference: CS\_WI\_BS005


Effective Date: 02Dec2019

Template No.:

#### 2.4. CHANGES TO ANALYSIS FROM PROTOCOL

- Change in definition of efficacy analysis set (EAS), in <u>section 4.4</u>.
- Analysis to be performed based on EAS has been revised to exclude PFS and OS in section 4.4.
- Subsequent oncology therapy was not defined in the protocol. The definition and analysis has been added in section 13 of SAP
- Changes on criteria of Hy's Law; "Serum AST or ALT ≥3 × ULN and ALP < 2x ULN and total bilirubin ≥2 × ULN" is changed to be "Hy's Law: Serum AST or ALT > 3 × ULN and ALP < 2x ULN and total bilirubin > 2 × ULN", in section 17.4.4.
- Changes on criteria of drug-induced liver injury (DILI); "Serum AST or ALT ≥3 × ULN together with total bilirubin ≥2 × ULN" is changed to be "Serum AST or ALT > 3 × ULN together with total bilirubin > 2 × ULN", in section 17.4.4.

#### 3. PLANNED ANALYSES

The timing of analysis for each cohort may be different depending on completion of each cohort, and the final analysis of the study will be conducted at the time of analysis of the last cohort. No formal interim analysis is planned for the study. However, the accrued data from any cohort may be analyzed for internal decision-making purposes; for example, to provide information for a future trial or external data disclosures. Then, the Database Lock (DBL) authorized by sponsor will be planned depending on the purpose of the analysis.

The final analysis will be planned to be carried out after a DBL. The DBL of final analysis is performed according to the study termination criteria (but not limited to) as below:

• The study is completed when all patients have discontinued study drug or the last enrolled patient have completed 1 year of treatment

OR

- If the study is terminated early for reasons including but not limited to:
  - The incidence or severity of adverse events (AEs) in this or other studies indicates a potential health hazard to patients.
  - o Patient enrollment is unsatisfactory.

#### 3.1. INTERIM ANALYSIS

No formal interim analysis is planned for the study. However, the accrued data from any cohort may be analyzed for internal decision-making purposes; for example, to provide information for a future trial or external data disclosures. During the analysis, selected summary for safety and anticancer activity of fruquintinib will be performed.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005



#### **3.2.** FINAL ANALYSIS

All final, planned analyses identified in this SAP will be performed by IQVIA Biostatistics following Sponsor Authorization of this Statistical Analysis Plan and Database Lock for this study.

#### 4. ANALYSIS SETS

Agreement and authorization of patients included/excluded from each analysis set will be conducted prior to database lock.

## 4.1. ALL PATIENTS ENROLLED SET [ENR]

The analysis set contains all patients who provide the informed consent form for this study.

# 4.2. SAFETY ANALYSIS SET [SAS] – (ALL TREATED POPULATION)

The analysis set includes all patients who have received at least one dose of fruquintinib. Patients in the SAS will be analyzed by their actual dose initially received. If patients have dose reduction during the study, all data will be summarized/analyzed on the initial dose of study drug received.

All safety analyses except for DLT summaries, along with PFS and OS will be based on the SAS.

If there is any doubt whether a patient was treated or not, they will be assumed treated for the purpose of analysis.

## 4.3. DOSE-LIMITING TOXICITY EVALUABLE SET [DLT]

The analysis set comprises all SAS patients who are evaluable for DLT assessment. DLT evaluable patients are identified if [Yes] is ticked as the response to "DLT Evaluable Patients" on CRF. DLT set and summaries will only apply to dose escalation phase.

## 4.4. EFFICACY ANALYSIS SET [EAS]

This analysis set includes all patients who have received at least 1 dose of fruquintinib, have a measurable lesion (target lesions ≥ 10 mm) at the baseline tumor assessment, and either (i) have had at least one post-baseline tumor assessment, or (ii) do not have post-dose tumor assessment but have clinical progression as noted by the investigator, or have died due to disease progression before their first post-baseline tumor scan. All efficacy endpoints (i.e. BOR, ORR, DCR, DoR, and best percentage change from baseline in tumor size), not including PFS and OS, will be summarized based on this analysis set.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

 Effective Date:
 02Dec2019



#### 5. GENERAL CONSIDERATIONS

#### 5.1. REFERENCE START DATE AND STUDY DAY

Reference start date is defined as the day of the first dose of study medication. Study Day will be calculated from the reference start date and will be used to show start/ stop day of assessments and events. Study day will appear in every listing where an assessment date or event date appears.

If the date of the event is on or after the reference date then:

Study Day = (date of event - reference date) + 1.

If the date of the event is prior to the reference date then:

Study Day = (date of event - reference date).

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings, but Study Day and any corresponding durations will be presented based on the imputations specified in <u>section</u> 6.3.

#### 5.2. BASELINE

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered baseline, unless additional information collected on eCRF indicate otherwise.

For example, ECG will be considered being performed post-baseline if assessment date coincides with the reference start date but "Time Point" on "ECG (ECG)" form indicates the assessment was performed "Post-dose 3 hours (± 15 minutes)". Adverse Events (AEs) onset on the reference start date and with "Did the adverse event occur prior to the start of study treatment?" in "Adverse Events (AE)" form answered as "No" or not being answered will be considered as post-baseline. Medications commencing the reference start date will be considered post-baseline.

#### 5.3. UNSCHEDULED VISITS AND EARLY TERMINATION DATA

In general, for by-visit summaries, data recorded at the nominal visit will be presented. Unscheduled measurements will not be included in by-visit summaries, but will contribute to the best/ worst case value where required (e.g., shift table).

Listings will include scheduled, unscheduled, and early discontinuation data.

Author:


Template No.: Reference: CS\_WI\_BS005

Effective Date: 02Dec2019

#### **5.4.** WINDOWING CONVENTIONS

The visit-window mapping is described in <u>APPENDIX 4</u>. Visit-based summaries will be based on the windowed visits. All data, whether or not within the visit windows, will be presented in listings.

For windowed visits during the treatment cycles,

- If more than 1 assessment occurs during a visit window, the assessment closest to the scheduled day will be assigned to the windowed visit.
- If two assessments are equidistant from the scheduled day, the later assessment will be assigned to the windowed visit.
- If there are multiple assessments on the same day, the worst case will be used.

For the post-treatment visit, the last assessment in the window will be included in the summary. The window for the post-treatment visit will be "from the last dose date + 8 days to the last dose date + 37 days".

For a patient who prematurely discontinues the study, the premature visit will be slotted accordingly.

#### 5.5. STATISTICAL TESTS

No formal statistical hypotheses will be tested in this study.

Two-sided 95% confidence intervals will be calculated and two-sided, unless otherwise specified in the description of the analyses.

#### **5.6.** COMMON CALCULATIONS

For quantitative measurements, change from baseline will be calculated as:

Test Value at Visit X – Baseline Value

#### 5.7. SOFTWARE VERSION

All analyses will be conducted with SAS version 9.4 or higher based on Enterprise Guide version 7.1.

#### 6. STATISTICAL CONSIDERATIONS

## 6.1. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

No adjustment will be performed.

Document:

Author:


18Feb2022

Template No.:

Reference: CS\_WI\_BS005

Effective Date: 02Dec2019

#### **6.2.** MULTICENTER STUDIES

This study is planned to be carried out at up to 10 sites. However, no adjustment in aspect of site effect will be performed. Data from all centers will be pooled for the analysis.

#### 6.3. MISSING DATA

Generally, the missing efficacy and safety data will not be imputed except for the critical missing and partial dates which will be handled as described in this section. In the situation where partial or missing date are imputed, the date will appear partial or missing in the listings, while imputed date will only be used for calculation.

#### 6.3.1. MISSING DATES INFORMATION OF STUDY TREATMENT

When the date of the last dose of study treatment is missing for a patient, all efforts should be made to obtain the date from the investigator. If it is still missing after all efforts, the last dose date collected from the [Study Drug Administration] page of or data cut-off date (if applicable) will be used in the calculation of treatment duration.

#### **6.3.2.** MISSING OR INCOMPLETE DATE INFORMATION FOR ADVERSE EVENT DATE

For the purpose of determining whether an adverse event (AE) is treatment emergent (see section 17.2.1), incomplete start dates and/or stop dates will be imputed. Start date will be imputed first when the start date and stop date are both incomplete for a patient. If the field of year is missing or start date of an AE is completely missing, then no value will be imputed. The following rules will be applied to impute the incomplete start date, assuming year is available.

#### Missing or incomplete start date

- In case the start date of an AE is in the same year as reference start date (when only year is recorded), or the start date is in the same month and year (if only the day is missing) as the reference start date, then the start date of the AE will be imputed by the reference start date or the AE resolution date, whichever occurs earlier.
- If the day and month parts of the AE onset date are missing and occur in the same year as the first dose of study drug, the date of the first dose of study drug will be used as the onset date of the AE. If an AE is observed on different year of first dose, January 1<sup>st</sup> will be used to complete the onset date of the AE.
- If only the day part of the AE onset date is missing and occurs in the same month and year as the first dose date of study drug, the date of first dose of study drug will be used as the onset date of the AE. Otherwise, the first day of the month will be used to complete the onset date of the AE.
- In all other cases, imputation will not be performed.

Here are some examples.

| Incomplete Date of Onset | Reference Start Date | Imputed Date |
|--------------------------|----------------------|---------------|
| (DD MMM YYYY) | (DD MMM YYYY) | (DD MMM YYYY) |
| | 10Apr2017 | |

Document:

Author:


Template No.:

Reference: CS\_WI\_BS005

Effective Date: 02Dec2019



| Incomplete Date of Onset | Reference Start Date | Imputed Date |
|--------------------------|----------------------|----------------------------|
| (DD MMM YYYY) | (DD MMM YYYY) | (DD MMM YYYY) |
| 2017 | 10Apr2017 | 10Apr2017 |
| 2018 | 10Apr2017 | 01Jan2018 (because the AE |
| | | onsets after the reference |
| | | date) |
| Apr2017 | 10Apr2017 | 10Apr2017 |
| Oct2017 | 10Apr2017 | 01Oct2017 |
| 052017 | 10Apr2017 | 052017 |

#### Missing or incomplete stop date

Incomplete stop dates will be imputed to the last possible date:

- If the known part(s) of the AE end date is (are) the same as the death date/ end of study date, the AE end date will be imputed by the death date/ end of study date, whichever occurs earlier.
- In all other cases, the AE end date will be imputed to the last day of the month if only the day is missing or imputed to with 31st December if both day and month are missing.
- If the imputed stop date is before the start date (imputed or non-imputed start date), then the stop date will be imputed using start date.
- If the end date is completely missing or the year part is unknown, the end date will not be imputed.

Here are some examples:

| Incomplete AE End Date | Date of Death/ End of Study | Imputed Date |
|---|---|---|
| (DD MMM YYYY) | (DD MMM YYYY) | (DD MMM YYYY) |
| May2017 | Not Available/ Not Available | 31May2017 |
| Sep2017 (known part the SAME as date of death/ end of study) | / 09Sep2017 | 09Sep2017 |
| 2017 (known part the SAME as date of death/ end of study) | 09Sep2017/ 09Sep2017 | 09Sep2017 |
| Jun2017 (known part DIFFERENT from date of death/ end of study) | 09Sep2017/ 09Sep2017 | 30Jun2017 |
| | / 09Sep2017 | |
| 31Dec | 09Sep2017/ 09Sep2017 | 31Dec |
| 2018 | 09Oct2019/ 09Oct2019 | 31Dec2018 |

 Document:
 2.5

 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005


## 6.3.3. MISSING OR INCOMPLETE DATE INFORMATION FOR CONCOMITANT MEDICATION/ PROCEDURE

The imputation rule is the same as described for adverse event.

## 6.3.4. MISSING OR INCOMPLETE DATE INFORMATION FOR PRIMARY DIAGNOSIS DATE AND METASTATIC DIAGNOSIS DATE

Imputation will only be applied in case the field of year is available. If year and month are known but the day is unknown, day will be imputed as 15. If only year is known, month and day will be imputed to July 1<sup>st</sup>. If the diagnosis date is completely missing or the year part is unknown, the diagnosis date will not be imputed.

#### 6.3.5. Missing or Incomplete Date Information for Efficacy Data

When a partial new anticancer therapy starting date is reported, every effort will be made to identify the precedence relationship of starting date of new anticancer therapy relative to last dosing date of study drug and the date of disease progression (if happened). According to the confirmed precedence relationship, partial new anticancer therapy date will be imputed to the earliest possible date:

- Day will be imputed as 1 if year and month are known; month and day will be imputed as Jan 1<sup>st</sup> if only year is known.
- In rare case, if year and month of death date are known but the day is unknown, day will be imputed as 15. For example, if a patient is reported to die on Dec2017, the death date will be imputed as 15 Dec2017.

However, the imputed anticancer start date will be adjusted based on corresponding date in different scenario as shown below, the imputed date will be set to the date according to which it will be adjusted if the originally imputed date is earlier than the corresponding date:

- Adjust based on the date of first dose in case that anticancer therapy starts earlier than both last dosing date and disease progression.
- Adjust based on the last dosing date/the date of disease progression which occurs earlier in case that anticancer therapy is initiated after last dosing date but before disease progression date or vice versa.
- Adjust based on the last dosing date/the date of disease progression which occurs later in case that anticancer therapy is initiated after both last dosing and disease progression.

#### **6.4.** MULTIPLE COMPARISONS/ MULTIPLICITY

There are no requirements for multiplicity adjustments in this study.

#### 6.5. EXAMINATION OF SUBGROUPS

No subgroup analyses will be performed for this study.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

 Effective Date: 02Dec2019
 02Dec2019



#### 7. OUTPUT PRESENTATIONS

Appendix 2 shows conventions for presentation of data in outputs.

Format and content of summary tables, figures, and listings are presented as mock shells for TFLs and provided by IQVIA Biostatistics.

Continuous variables will be summarized using descriptive statistics including, number of patients (n), mean, median, standard deviation (STD), 25% and 75% quantiles, minimum and maximum. Categorical variables will be summarized with number and percentage and presented in frequency tables. All results will be presented by dose cohort (only in dose escalation phase) or tumor specific cohorts (only in dose expansion phase).

Qualitative variables will be summarized by count(s) and percentages (%).

Percentages will be reported with 1 decimal point; if the count is 0, no percentage will be presented. Value of percentage less than 1% will be presented as "<1%." Value of percentage less than 100% but >99% will be presented as ">99%." Any rounding will be done after all calculations are made.

#### 8. DISPOSITION AND WITHDRAWALS

#### 8.1. ENROLLMENT

Information of all patients who provided informed consent (that is the ENR) will be included in the summary of disposition and withdrawals for this study. A summary table will be generated to provide the following:

- Number of patients who signed the informed consent
- Number of screen failures
- Reason for screen failure
- Number of patients who passed screening
- Number of patients who withdrew consent before study treatment
- Number of patients who received treatment

A separate table will be presented to show the patients included in each analysis set and reason for exclusion from an analysis set.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

 Effective Date: 02Dec2019
 02Dec2019




# 8.2. PATIENT STATUS AT TREATMENT AND STUDY COMPLETION

Patient status at treatment and study completion will be listed and summarized for SAS. The listing will include individual information (i.e. site and patient number, informed consent information), whether patients discontinued from the treatment and the reasons for the discontinuation, along with the date of first/ last dose, duration of treatment, and the date of discontinuation from the treatment. The same information will be provided for patients who discontinued from the study. The following summaries will be presented:

- Patients still on treatment
- Reason for study drug discontinuation (for study drug)
- Number of patients going into Survival follow-up
- Number and percentage of patients who discontinue the study
- Reason for study discontinuation

A flowchart for disposition will be presented.

#### 9. PROTOCOL DEVIATION

Protocol deviations are recorded as critical, major or minor in Clinical Trial Management System (CTMS) and are classified into 10 categories:

- Administrative Criteria
- Eligibility and Entry Criteria
- Informed Consent Criteria
- IP Compliance
- Laboratory Assessment Criteria
- Regulatory or Ethics Approvals Criteria
- Serious Adverse Event Criteria
- Study Procedures Criteria
- Visit Schedule Criteria
- Other Criteria

Major protocol deviations are those recorded as critical or major.

All subject-level protocol deviations will be presented in listing including deviation date and severity.

| Document: | | |
|--------------|---------------|------------------------|
| Template No | o.: | Reference: CS_WI_BS005 |
| Effective Da | te: 02Dec2019 | |



#### 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented for the SAS. Data listing will also be provided.

No statistical testing will be carried out for demographic or other baseline characteristics.

The following demographic and other baseline characteristics will be reported for this study:

- Age (years) calculated relative to date of consent; summarized as both continuous variable and categorical variable (< 65 vs. ≥ 65 years)</li>
- Gender
- Race
- Ethnicity
- Weight (kg)
- Height (cm)
- BMI (kg/m²): summarized as both continuous and categorical variable (<18.5, ≥18.5 and <24, ≥24 kg/m²)</li>
- Baseline ECOG performance status (0, 1, 2, 3, 4, 5)

#### 10.1. DERIVATIONS

BMI  $(kg/m^2)$  = weight (kg)/ height  $(m)^2$ 

#### 11. SURGICAL AND MEDICAL HISTORY

Medical and surgical history will be coded by MedDRA Version 23.1 or higher and summarized separately for SAS; results will be expressed by system organ class (SOC) and preferred term (PT) in descending order of the frequency in total. For SOCs or PTs with the same frequency, results will be sorted alphabetically. Individual patient listings of and medical/surgical history will also be provided for the SAS.

#### 12. ONCOLOGY HISTORY

Oncology history information will be presented for the SAS. The following oncology history information will be summarized:

Document:

Author:


Template No.:

Reference: CS\_WI\_BS005


- Primary diagnosis of malignancy
- Time since primary diagnosis to first dose of study treatment (months)
- Primary site
- Diagnosis of malignancy at enrollment
- Metastatic status (yes, no)
- Number of metastatic sites: both continuous variable and categorical variable  $(0, 1, 2, \ge 3)$
- Time since first metastasis diagnosis to first dose of study treatment (months)
- TNM stage at enrollment
- Disease stage at enrollment
- Histological classification at enrollment (Adenocarcinoma, Adenosquamous Carcinoma, Carcinoid, Clear Cell Carcinoma, Indeterminate, Sarcoma, Squamous (except squamous non-small cell lung cancer [NSCLC], Other)
- Prior use of VEGF-R inhibitor (yes, no)
- Prior use of VEGF inhibitor (yes, no)
- Time since last systemic anti-neoplastic therapies to first dose of study treatment (months)
- Liver metastasis (yes, no): obtained based on whether the liver organ was involved in the target and non-target lesion tumor scan assessment at the baseline.

#### 12.1. **DERIVATIONS**

- Time since primary diagnosis to first dose of study treatment (months) = (Date of first dose of study treatment Date of primary diagnosis)/30.4375
- Time since first metastasis diagnosis to first dose date (months) = (Date of first dose of study treatment Date of first metastasis diagnosis)/ 30.4375
- Time since last systemic anti-neoplastic therapies to first dose of study treatment (months) = (Date of first dose of study treatment Date of last systemic anti-neoplastic therapies)/ 30.4375

#### 13. ONCOLOGICAL THERAPIES

#### 13.1. PRIOR ONCOLOGICAL THERAPY

Prior oncological therapy information are recorded as following: Prior oncology medication information, Prior oncology radiotherapy information, Prior oncology surgery and procedure information.

Prior oncology medication will be coded using World Health Organization Drug Dictionary Enhanced (WHO DDE) Version SEP2020. Prior oncology surgery and procedures will be coded using MedDRA Version 23.1 or higher.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

 Effective Date: 02Dec2019
 02Dec2019

Prior oncology medications will be presented by Anatomical Therapeutic Classification (ATC)-2<sup>nd</sup>-level term (ATC level 2) and by PTs for each dose and/ or disease cohort in each phase. ATC class and PT will be sorted in descending frequency of the total number of patients with at least one condition in the corresponding category; ATCs/PTs will be presented alphabetically for ATCs/PTs of the same total frequency. In addition, number and percent of patients who have received prior oncology medication, regimen number, and category of regimen number will be summarized for prior oncology medication.

Prior oncology surgery and procedures will be presented by SOC and PT for each cohort in each phase. SOC and PT will be sorted in descending frequency of the total number of patients with at least one condition in the corresponding category, SOCs/PTs will be presented alphabetically for SOCs/PTs of the same total frequency. Corresponding listings will be provided.

### 13.2. SUBSEQUENT ONCOLOGY THERAPY

Subsequent oncology therapies taken after end of treatment will be collected in below forms:

- "Oncology Medication (CHEMO1)"
- "Oncology Radiotherapy"
- "Oncology Surgery and Procedure"

Subsequent oncology therapies are defined as therapies started after the last dose of study medication. The following information will be summarized and listed for subsequent therapy:

- Number of subsequent oncology medications
- Number of subsequent regimen
- Category of number of subsequent regimen

Subsequent oncology (or anti-tumor) medications will also be presented by ATC level 2 and by PTs for each dose/disease cohort in each phase.

Subsequent anti-tumor therapy will be flagged in the listing of oncology medication/ radiotherapy/ surgery.

### 14. MEDICATIONS AND PROCEDURES

Medications and procedures information are recorded as following:

- Prior and concomitant medication information
- Prior and concomitant procedure information

| Document: | |
|---------------------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |
| Effective Date: 02Dec2019 | |

'Prior' medications/procedures are medications/procedures which started prior to the first dose of study medication.

'Concomitant' medications/procedures except for oncology therapies are medications which ended on or after the date of first dose of study medication or were ongoing at the end of the study, and start no later than 37 days following last dose administration.

A medication may be both prior and concomitant if it meets 2 above-mentioned definitions.

#### 14.1. Prior and Concomitant Medication

Medications will be coded using World Health Organization Drug Dictionary Enhanced (WHO DDE), Versions SEP2020 or higher. See <u>section 6.3.3</u> for handling of partial dates for medications, in the case where it is not possible to define a medication as prior and concomitant, the medication will be classified by the worst case, i.e. concomitant.

Concomitant medications will be presented by ATC level 2 and by PTs for each dose and/ or disease cohort in each phase. ATC class and PT will be sorted in descending frequency of the total number of patients with at least one condition in the corresponding category, ATCs/PTs will be presented alphabetically for ATCs/PTs of the same total frequency.

Prior and concomitant medications will be presented in listings with flag to differentiate whether the medication is prior medication or concomitant medication.

#### 14.2. CONCOMITANT PROCEDURES

Surgery and procedures will be coded using MedDRA Version 23.1 or higher. Concomitant procedures will be presented by SOC and PT for each dose and/ or disease cohort in each phase.

SOC and PT will be sorted in descending frequency of the total number of patients with at least one condition in the corresponding category, SOCs/PTs will be presented alphabetically for SOCs/PTs of the same total frequency. Prior and concomitant surgery will be listed and flagged like the listing of prior and concomitant medication.

#### 15. STUDY MEDICATION EXPOSURE

Exposure to study medication and compliance will be presented for the SAS.

The planned treatment is given at either 3mg QD or 5mg QD in the corresponding study phase and dose and/ or disease cohort. In each 28-day cycle, a patient will take medication in the first 3 weeks followed by 1 week off treatment. Study drug administration and derived exposure information will be summarized and listed.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

 Effective Date: 02Dec2019
 02Dec2019



#### 15.1. EXPOSURE TO STUDY MEDICATION

Below variables will be summarized:

- Number of cycle(s) received: the number of cycles in which at least one dose of Fruquintinib or placebo is taken. The number of cycles could be further categorized into:
  - $\circ$  1, 2, 3, 4, 5, 6 and > 6
- Total duration of exposure (days)
- Cumulative dose (mg)
- Dose intensity (mg/day)
- Relative dose intensity (RDI, %): both continuous variable and categorical variable (< 50%; 50 < 70%; 70 < 90%; 90 < 110%;  $\ge 110\%$ )
- Actual duration of study treatment (days)
- Percentage intended dose (PID)
- Number of patients with any dose modification (including both drug interruption, dose increase, and dose reduction)
- Frequency of dose modification: 0, 1, 2, 3, 4, 5, 6, >6
- Number of patients experienced drug interruption
- Frequency of drug interruptions:  $0, 1, \ge 2$
- Number of patients with any dose reduction
- Reduction from 5mg to 4mg
- Reduction from 4mg to 3mg
- Frequency of dose reduction: 0, 1, 2

#### 15.2. STUDY MEDICATION COMPLIANCE

The study medication compliance is quantified with relative dose (RD, %) of study medication. RD is calculated as the cumulative dose taken divided by the planned total dose in the corresponding period, expressed as a percentage, see <a href="section 15.3">section 15.3</a> for more details. RDI (%) and RD (%) will be categorized as stated above in <a href="Section 15.1">Section 15.1</a>.

#### 15.3. DERIVATIONS

- Total duration of exposure (days) is calculated from the first dose date of study drug in Cycle 1 to the last dose date of study drug + 8 days or death date, whichever comes earlier if treatment is discontinued, or to the cut-off date. if treatment is still ongoing.
- Actual duration of exposure (days) = Sum of the days with study drug administered

Algorithms for calculating parameters relevant to the dose exposure and intensity are listed in Table below:




| Parameter | Description/ Formula [a] |
|---|---|
| Dosing schedule per | 5 mg PO QD between Days 1 and Day 21, followed by 1-week off |
| protocol# | |
| Cumulative dose (mg) [b] | $\sum$ [5 × (all dispensed 5-mg tablets – total returned 5-mg tablets - total lost 5-mg |
| | tablets in a cycle) + 1 × (all dispensed 1-mg tablets – total returned 1-mg tablets |
| | - total lost 1-mg tablets in a cycle)] |
| Dose intensity (mg/day) | Cumulative dose (mg) / Total duration of exposure (day) |
| Relative dose intensity | 100 * [Dose intensity (mg/day) / (5 × 21/28, mg/day)] |
| (RDI, %) # | |
| Relative Dose (RD, %)# | 100 * [Cumulative dose (mg) / (5 × 21 × number of cycles received (mg)] |
| Percentage intended dose | 100 * [(total number of days with any recorded doses) / total duration of |
| (PID, %) [c] | exposure (days)] |

<sup>[</sup>a]In the study, there are the other dose level of "3mg QD" used.

[c]Given the dose schedule of a 4-week cycle in the protocol, 3 weeks on/ 1 week off, the reference value is 0.75.

#### 16. EFFICACY OUTCOMES

Analyses of efficacy outcomes are based on EAS except PFS and OS, which are estimated based on SAS.

## 16.1. PRIMARY EFFICACY VARIABLE(S) & DERIVATION(S)

#### 16.1.1. BEST OVERALL RESPONSE (BOR)

BOR will be determined using time point responses (TPRs) up until the last evaluable TPR prior to or on the date of (i) disease progression as defined by RECIST Version 1.1 (Eisenhauer et al., 2009) or death; or (ii) withdrawal of consent; or (iii) receiving subsequent anti-cancer therapy, whichever is earlier.

The timing of an overall TPR will always be derived based on scan dates not response assessment dates. For a scheduled tumor scan assessment, it is expected that there may be a variation for the actual timing of scans among target, non-target, and new lesions. In assigning a date for the overall response assessment at a visit, the earliest date collected at that visit will be used. Within a grouped timepoint, if there are multiple assessments on different dates for the same target lesions, the last assessment will be used.

A patient's BOR will be determined based on APPENDIX 3.

| Document: | |
|---------------------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |
| Effective Date: 02Dec2019 | |

<sup>[</sup>b]In the study, both 1-mg and 5-mg fruquintinib are provided for oral administration. When dose adjustment is required, 1-mg fruquintinib is always used. Before calculating the cumulative dose, total number of 1-mg and 5-mg tablets taken should be counted separately.

<sup>#</sup> indicates 5 (mg) should be replaced with 3 (mg) for calculation in Cohort "3 mg QD".


There are two ways of assigning BOR for a patient when the minimum interval for confirmation of CR and PR is not satisfied or if there are no confirmatory scans for CR and PR:

- Adding two more response categories as: unconfirmed CR, unconfirmed PR.
- Assigning BOR as SD, that is, both the unconfirmed CR and unconfirmed PR will be SD.

Both ways of assigning BOR will be implemented.

The number and percentage of patients in each category of derived BOR (Confirmed CR, Confirmed PR, SD, PD, or NE) will be summarized.

#### 16.1.2. OBJECTIVE RESPONSE RATE (ORR)

Objective response rate (ORR) will be calculated using two different ways:

- Scenario #1: ORR will be calculated using a strict interpretation of RECIST Version 1.1. Objective response will be derived as no/yes variable. Patients with a BOR of confirmed CR or PR will be assigned 'Yes'. Patients not having a BOR of confirmed CR or PR will be assigned 'No'. Hence, ORR is defined as the proportion of patients with objective response being "Yes".
- Scenario #2: ORR<sub>UNCONFIRMED</sub> will be calculated using all responses regardless of confirmation. Objective response will be derived as no/yes variable. Patients with a BOR of confirmed CR, confirmed PR, unconfirmed CR or unconfirmed PR will be assigned "Yes". All patients with other BOR values will be assigned "No". Hence, ORR<sub>UNCONFIRMED</sub> is defined as the proportion of patients with objective response being "Yes".

#### 16.1.3. DURATION OF RESPONSE (DOR)

The DoR is defined as the time from the date of the first objective response (CR or PR which is subsequently confirmed) until the date of the documented progression or of death, whichever comes first. DoR will only be analyzed for patients whose BOR is either CR or PR. Censoring will follow the rules outlined below for PFS in Section 16.1.5.

#### 16.1.4. DURATION CONTROL RATE (DCR)

The DCR is defined as the percentage of patients in EAS with a BOR of confirmed CR, confirmed PR or SD for 7 weeks.

#### 16.1.5. PROGRESSION FREE SURVIVAL (PFS)

The PFS is defined as the time from date of first dosing until the date of an objective disease progression as defined by RECIST Version 1.1 (Eisenhauer et al., 2009) or death due to any cause, whichever comes first. More specifically, PFS will be determined using all the assessment data up until the last evaluable visit prior to or on

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

 Effective Date: 02Dec2019
 02Dec2019


the date of (i) disease progression as defined by RECIST Version 1.1 or death; or (ii) withdrawal of consent; or (iii) receiving subsequent anti-cancer therapy, whichever is earlier.

The rule of censoring/ event is summarized in Table 1.

The PFS time will always be derived based on scan dates not tumor assessment dates. If PD is documented between scheduled visits, the actual date of documented progression will be used as an uncensored value in the analysis of PFS.

RECIST assessments/scans contributing towards a particular visit may be performed on different dates. The following rules will be applied:

- Date of progression will be determined based on the earliest of the dates of the component that triggered the progression.
- When censoring a patient for PFS the patient will be censored at the latest of the dates contributing to a particular overall visit assessment.

Table 1 Progression free survival

| Description | Event/ | Date of Event/Censor |
|---|---|---|
| | Censor | |
| Documented progression before starting use of | Event | Date of first documented disease progression |
| new anticancer treatment and without missing | | |
| two consecutive tumor assessment visits | | |
| Death without progression | Event | Date of death |
| Progression or death after two or more | Censor | Date of last adequate tumor assessment before |
| consecutive missed tumor assessments | | two consecutive missed tumor assessment visits |
| No evaluable baseline tumor assessment | Censor | Date of first dosing of study treatment |
| No evaluable tumor assessment after first dose | Censor | Date of first dosing of study treatment |
| of study treatment | | |
| New anticancer treatment started prior to | Censor | Date of last evaluable tumor assessment before |
| documented disease progression or death on | | start use of new anticancer treatment/two |
| study | | consecutive missed tumor assessment visits |
| No progression and no death before end of | Censor | Date of last evaluable tumor assessment |
| study or data cut-off | | |

Note: An adequate radiologic assessment is defined as an assessment where the Investigator determined radiological response is CR, PR, SD, or PD. If PD and new anti-cancer therapy occur on the same day, will assume that the progression was documented first, e.g. outcome is progression and the date is the date of the assessment of progression.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005


Note: Two consecutive scheduled tumor assessments is equal to 126 days (=2\* (8 weeks \*7+ 7 days)) since previous evaluable RECIST 1.1 or baseline assessment if there is no post baseline tumor assessment.

#### 16.1.6. OVERALL SURVIVAL (OS)

The OS (in months) refers to the time interval between the first dose date and the date of death (any cause). The last known alive date (i.e. the last follow-up date in patients on study or the date of EOS in patients withdrawn from the study) will be used as the censoring date for patients who have not died at the time of the statistical analysis. Patients lacking data beyond the first dose date will have their survival time censored at the first dose date.

#### 16.1.7. TUMOR SHRINKAGE

Tumor shrinkage will be estimated using data on sum of diameters of target lesion based on EAS. Percentage change in tumor size will be determined for patients with measurable disease at baseline and will be derived for each tumor assessment.

## **16.2.** ANALYSIS OF EFFICACY VARIABLE(S)

The efficacy endpoints include ORR, DCR, DoR, PFS and OS. Efficacy data will be listed and summarized by dose cohort (only in dose escalation phase) or tumor specific cohorts (only in dose expansion phase) and disease type if applicable.

#### ORR, DCR, and DoR

The ORR and DCR will be summarized with percentages and 95% exact Clopper-Pearson confidence interval based on EAS.

DOR will be summarized using Kaplan-Meier method, and the descriptive statistics of median, 25% and 75% percentiles along with their 95% CIs will be calculated. It will be based on the EAS. The supportive data listings will also be provided.

#### PFS. OS. and Duration to Follow-Un

PFS and OS will be similarly summarized as DOR, and in addition to the quartile summary from Kaplan-Meier method, Kaplan-Meier estimates will be provided for the rates at 12, 16, 20, and 24 weeks along with their 95% CIs based on the Brookmeyer and Crowley method (1982).

In addition, duration (months) to follow-up for overall survival would be summarized by Kaplan-Meier method. Duration to follow-up refers to the time interval between date of first study drug administration and last date known to be alive for subjects who have not yet been reported to have died by the time of analysis, i.e. (date of last known to be alive – date of first study drug administration  $\pm 1$ )/ 30.475. Subjects who are reported to have died would be censored at death date.

#### **Tumor Shrinkage**

Document:

Author:


Template No.:

Reference: CS\_WI\_BS005


Percentage change in tumor size from baseline will be determined for patients with measurable disease at baseline and derived at each visit by the percentage change in the sum of the diameters of target lesions (TLs) compared to baseline. Best (minimum) percentage change from baseline (PCFB) in tumor size will be summarized using descriptive statistics and a waterfall plot will be presented also. Best post-baseline sum of diameter is defined as the sum of diameter with either the largest decrease or smallest increase from baseline sum of diameter at a single post-baseline evaluable tumor assessment visit before RECIST progression of disease. More details please refer to section 16.1.7.

#### 17. SAFETY OUTCOMES

Unless otherwise specified, the overall safety evaluation period is from the first date of study drug administration to no later than 37 days after the date of last study treatment administration. All outputs for safety outcomes will be based on the SAS.

There will be no statistical comparisons between the treatment groups for safety data, unless otherwise specified with the relevant section.

Safety will be assessed through summaries of adverse events, changes in laboratory test results, changes in vital signs and change in ECG. Safety data will be listed and summarized. Incidence of DLTs will be listed by dose cohort for dose escalation phase only.

#### 17.1. DLTs

A DLT is defined as one of the following toxicities occurring during the DLT assessment window (Cycle 1) and determined by the investigator to have a reasonable possibility of being related to fruquintinib. All DLT analysis will be performed for dose escalation phase only. In addition to summarizing the proportion of patients with DLTs, the DLT categories will also be summarized as follows:

- Any Grade 4 non-hematologic toxicity;
- Any Grade 3 non-hematologic toxicity related to study drug except for nausea/vomiting, diarrhea, constipation, hypertension and electrolyte imbalances downgraded within 3 days with appropriate supportive treatment;
- Grade 4 neutropenia lasting > 3 days;
- Grade 3 febrile neutropenia (absolute neutrophil count < 1.0 x 109/L with a single temperature of > 38.3 °C or a sustained temperature of ≥38 °C for more than 1 hour;
- Grade 4 thrombocytopenia or Grade 3 thrombocytopenia associated with bleeding;
- DLT leading to dose interruption for > 14 days due to toxicity

The individual data of DLTs will also be listed by dose and/ or disease cohort and by patient.

| Document: | |
|---------------------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |
| Effective Date: 02Dec2019 | |

#### 17.2. ADVERSE EVENTS

AEs will be coded using Medical Dictionary for Drug Regulatory Activities (MedDRA) central coding dictionary, Version 23.1 or higher.

Treatment emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity on or after the first dose of study medication and no later than 37 days after the date of last study treatment. In case that the AE onset date coincide with the first dose date of study treatment, AE will be considered as TEAE if the response of question "Did the adverse event occur prior to the start of study treatment?" in AE form is "No".

See <u>section 6.3.2</u> for handling of partial dates for AEs. In the case where it is not possible to define an AE as treatment emergent or not, (i.e., the required imputed dates are missing or partial) the AE will be classified by the worst case, i.e. treatment emergent.

An overall summary of number of patients within each of the categories described in the sub-section below, will be provided.

Listings will include all the AEs being reported during the study with flag to distinguish TEAEs and Non-TEAEs. Imputed AE dates will not be presented in the listings.

#### **17.2.1. ALL TEAES**

Incidence of TEAEs will be presented by System Organ Class (SOC) and Preferred Term (PT) and also broken down further by maximum severity for each phase, each dose and disease cohort and overall. The study drug related TEAEs will also be summarized in the similar way.

#### 17.2.1.1. Severity

Effective Date: 02Dec2019

AE severity will be graded to 5 grades (Grade 1 to Grade 5) according to the national cancer institute common terminology criteria for adverse event (NCI CTCAE) V4.03.

TEAEs starting after the first dose of study medication with a missing severity will be classified as Grade 3. If a patient reports a TEAE more than once within that SOC/ PT, the AE with the worst-case severity will be used in the corresponding severity summaries. A summary table for TEAE with grade >= 3 will also be presented by dose or disease cohort.

#### 17.2.1.2. Relationship to Study Drug

The relationship, as indicated by investigator, is classed as "Unrelated" and "Related". A study drug "related" TEAE is defined as a TEAE with response of "Yes" to the field "Possible causality to study drug?" on the "Adverse Event (AE)" form of the eCRF. TEAEs with a missing causality to study drug will be regarded as "Related" to study drug. If a patient reports the same AE more than once within that SOC/ PT, the AE with the worst case relationship to study drug will be used in the corresponding relationship summaries.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005



#### 17.2.2. TEAES LEADING TO DOSE INTERRUPTION OR REDUCTION

TEAEs leading to dose interruption or reduction will be identified as those TEAEs with a response of either "Drug Interrupted" or "Dose Reduced".

For TEAEs leading to dose interruption or reduction, summaries of incidence rates (frequencies and percentages) by SOC and PT will be prepared. Summaries for TEAEs leading to dose interruption or reduction by SOC and PT will be further limited to study medication-related TEAE and broken down by maximum severity.

#### 17.2.3. TEAES LEADING TO DISCONTINUATION OF STUDY DRUG

TEAEs leading to permanent discontinuation of study drug will be identified as those TEAEs with a response of "Drug Withdrawal".

For TEAEs leading to discontinuation of study drug, summaries of incidence rates (frequencies and percentages) by SOC and PT will be prepared. Summaries for TEAEs leading to discontinuation of study drug by SOC and PT will be further broken down by maximum severity and strongest relationship to study drug.

TEAEs leading to discontinuation of study drug will also be listed.

#### 17.2.4. SERIOUS ADVERSE EVENTS

Serious adverse events (SAEs) are those events recorded with a response of "Yes" for the field "Is the adverse event serious?" on the "Adverse Events (AE)" form of eCRF. A summary of serious TEAEs by SOC and PT will be prepared. In addition, summaries for serious TEAEs by SOC and PT will be further broken down by maximum severity.

Listing of serious TEAE will also be provided.

#### 17.2.5. ADVERSE EVENTS LEADING TO DEATH

TEAEs leading to Death are those events with response of "Fatal. A summary of TEAEs leading to death by SOC and PT will be prepared.

TEAEs leading to death will also be listed.

#### 17.2.6. ADVERSE EVENTS OF SPECIAL INTEREST (AESI)

According to the IB Version 13.0 (dated 08 November 2021), treatment emergent adverse events of special interest (TEAESI) for fruquintinib are defined to include 10 categories:

- hepatic function abnormal
- haemorrhages
- hypertension
- infections
- thyroid dysfunction
- proteinuria
- dermatological toxicity
- gastrointestinal perforation

| Document: | |
|---------------------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |
| Effective Date: 02Dec2019 | |
- embolic and thrombotic events
- left ventricular ejection fraction decreased

The MedDRA terms used to define AESIs categories are listed in Table 2, for AESI categories (i.e. "haemorrhages", "hepatic function abnormal", "hypertension", "proteinuria", "thyroid dysfunction", "embolic and thrombotic events" "gastrointestinal perforation" and "left ventricular ejection fraction decreased"), the PTs to be included in these AESI categories are included in <u>Appendix 5</u>. These terms were selected by subjecting standardized MedDRA queries (SMQ) lists (narrow and/or broad scope depending on the category) for each category and had been used in the fruquintinib clinical development program for pharmacovigilance. TEAESI will be summarized by AESI category and PTs. Incidence rates (frequencies and percentages) will be presented by treatment arm. Similar by severity and by relationship summary tables will also be provided separately.

Table 2: MedDRA Terms Used for Adverse Events of Special Interest

| AESIs Category | Search terms/strategy |
|---|---|
| Dermatological toxicity | MedDRA SOC "skin and subcutaneous tissue disorders" |
| Hypertension | MedDRA SMQ "hypertension" (narrow) |
| Thyroid dysfunction | MedDRA SMQ "thyroid dysfunction" (broad) |
| Proteinuria | MedDRA SMQ "proteinuria" (narrow) |
| Hepatic function abnormal | MedDRA SMQ "drug related hepatic disorders-comprehensive |
| | search" (narrow) |
| Haemorrhages | MedDRA SMQ "haemorrhages" (narrow) |
| Infections | MedDRA SOC "infections and infestations" |
| Embolic and thrombotic events | MedDRA SMQ "embolic and thrombotic events" (narrow) |
| Gastrointestinal perforation | MedDRA SMQ "gastrointestinal perforation" (narrow) |
| Left ventricular ejection fraction decreased | MedDRA SMQ "cardiac failure" (narrow) |

Time to first TEAESI will also be summarized by AESI category for each dose and/ or disease cohort in each study phase. Time to first TEAESI is defined as time interval from date of first administration of study treatment to the earliest onset date among TEAEs within the same AESI categories. That is, if a patient has multiple AEs occurrences under the same AESI category, the earliest AE onset date will be used as the first onset date to the AESI category.

## **17.3. DEATHS**

Data on death will be listed, along with results of total number of patients died and cause of death summarized. Result of patients with on-study death, which is defined as the death after the first dose until 37 days after last dose, will also be tabulated. On-treatment death will be flagged.

## 17.4. LABORATORY EVALUATIONS

Results from the local laboratory will be included in the reporting of this study for Hematology, Serum chemistry, Coagulation, Urinalysis, 24-hours urine protein, and Thyroid function test.



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Indexes collected for laboratory assessments are shown in table below:

| Laboratory Test | Parameters |
|---|---|
| Hematology | red blood cell [RBC] count, hemoglobin, platelet count, white blood cell [WBC], |
| | neutrophils, lymphocytes, monocytes, eosinophils, basophils, hematocrit, |
| | reticulocyte count |
| Coagulation | activated partial thromboplastin time [aPTT], international normalized ratio [INR] |
| Serum chemistry | total protein, albumin, glucose, blood urea nitrogen [BUN], creatinine, creatinine |
| | clearance, alkaline phosphatase [ALP], lactate dehydrogenase [LDH], total |
| | bilirubin, Aspartate Aminotransferase [AST], Alanine Aminotransferase [ALT], |
| | calcium, magnesium, potassium, sodium, chloride, total cholesterol, triglycerides, |
| | uric acid, bicarbonate, phosphorus |
| Urinalysis | pH, glucose, protein, and blood |
| Thyroid function | thyroid stimulating hormone [TSH], free T3, and free T4 |

The non-protocol specified tests and urinalysis results will not be summarized; they will only be included in listings. Data recorded by the laboratory will be converted to the International System of Units (SI) and all presentations will use SI units. Quantitative laboratory measurements reported as "< X", i.e., below the lower limit of quantification (LLQ), or "> X", i.e., above the upper limit of quantification (ULQ), will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, i.e., as "< X" or "> X" in the listings. Quantitative data collected between after date of ICF and up to 37 days following the last dose of study medication will be used for analysis. The following summaries will be provided for laboratory data:

- Observed value and change from baseline by visit (for quantitative measurements)
- Shift from baseline to worst post-baseline CTCAE toxicity for laboratory abnormalities
- Shift from baseline to the worst post-baseline investigators' assessment (i.e., normal, abnormal but not clinically significant [NCS], abnormal and clinically significant [CS] for quantitative measurements and categorical measurements)

Both the scheduled and unscheduled assessments will be used to identify the worst post-baseline values. Listing of all laboratory data by patients, abnormal values identified according to normal range (low, normal and high) by programming and markedly abnormal criteria by investigators' assessment will be flagged.

#### 17.4.1. LABORATORY SPECIFIC DERIVATIONS

The SI unit conversion and CTCAE grade will be derived through programming.

| Document: | |
|---------------------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |
| Effective Date: 02Dec2019 | |

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

## 17.4.2. CTCAE GRADING FOR LABORATORY DATA

To identify laboratory values of potential clinical importance, laboratory results will be graded according to NCI CTCAE Ver. 4.03, where applicable (<u>APPENDIX 6</u>). All grading will be based on laboratory values (being direct or some derived, corrected values) only, regardless of its interventional or symptomatic consequences. Some modifications to the grading system will be applied:

- Grade 5 refers to fatal outcomes, which cannot be determined solely by laboratory values, therefore will not appear in the grading system.
- A further category denoted Grade 0 would include all laboratory values within normal range except missing values.
- Missing results shall be graded as missing.
- For some specific parameters with CTCAE grading in both high and low direction (e.g., calcium, glucose, magnesium, potassium, sodium), CTCAE in hyper and hypo directions will be presented separately, i.e., hyper for higher values of concern and hypo for lower values of concern.

Any graded abnormality that occurs following the initiation of study drug and represents at least a 1-grade change (i.e. increase or decrease) from the baseline assessment is defined as treatment emergent. The treatment-emergent laboratory abnormality defined by CTCAE will be summarized by CTCAE term, CTCAE toxicity grade, and visit. Any occurrence of grade 3 or grade 4 laboratory abnormality during the treatment period will also be summarized by visit.

#### 17.4.3. LABORATORY REFERENCE RANGES

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges in SI units and categorized as:

- Low: Below the lower limit of the laboratory reference range
- Normal: Within the laboratory reference range (upper and lower limit included)
- High: Above the upper limit of the laboratory reference range

#### 17.4.4. POTENTIAL DRUG-INDUCED LIVER INJURY (DILI)

Below events will be identified via programming and summarized by categories and dose and/ or disease cohort for the SAS. Separate listings for patients with DILI, as defined below, will also be provided.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005


- Hy's Law: Serum AST or ALT >3 × ULN and ALP < 2x ULN and total bilirubin >2 × ULN
- POTENTIAL DRUG-INDUCED LIVER INJURY (DILI): Serum AST or ALT >3 × ULN and total bilirubin >2 × ULN
- AST:
- $\circ$  > 3x ULN and < 5 x ULN.
- $> 5 \text{ x ULN and} \le 8 \text{ x ULN}$ ,
- $\circ$  > 8 x ULN and  $\leq$  10 x ULN,
- $> 10 \text{ x ULN and} \le 20 \text{ x ULN}$ ,
- $\circ$  > 20x ULN,
- AST>5x ULN for more than 5 weeks
- ALT:
- $\circ$  > 3x ULN and  $\leq$  5 x ULN,
- $> 5 \text{ x ULN and} \le 8 \text{ x ULN}$ ,
- $> 8 \times ULN \text{ and } \le 10 \times ULN,$
- $> 10 \text{ x ULN and } \le 20 \text{ x ULN},$
- $\circ$  > 20x ULN,
- $\circ$  > 5x ULN for more than 5 weeks

Lab abnormalities meeting the biochemical criteria for Hy's law is associated with a markedly increased possibility of severe DILI. These components will also be listed separately:

- ALP  $< 2 \times ULN$
- Total Bilirubin:
- $\circ$  >1.5 and < 2 x ULN
- $o > 2 \times ULN$

## 17.5. ECG EVALUATIONS

Results of the Electrocardiogram (ECG) will be included in the reporting of this study. Overall assessment of ECG up to 37 days following the date of last dose of study medication will be included for analysis.

The following ECG parameters will be reported for this study:

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

- Heart Rate (bpm)
- PR Interval (msec)
- QT Interval (msec)
- ORS Interval (msec)
- RR Interval (msec)
- QTcF Interval (msec)

Overall assessment of ECG (Investigator's judgment): Normal, NCS, CS.

The following summaries will be provided for ECG data:

- Observed and change from baseline by visit
- Markedly abnormal value and change of ECG by visit
- Shift table of change from baseline to worst post-baseline ECG assessment by investigator

Listing of ECG data (Assessment date, Timepoint, HR, PR interval, QT interval, QRS interval, RR interval, QTcF interval) by patients, with results which meet the markedly abnormal criteria being flagged.

#### 17.5.1. ECG SPECIFIC DERIVATIONS

QTcF values will be derived from the QT and RR intervals based on the formula of

$$QTcF = \frac{QT}{\sqrt[3]{RR}},$$

If QT and/or RR is missing, the QTcF will be left as missing.

#### 17.5.2. MARKEDLY ABNORMAL CRITERIA

Markedly abnormal criteria for ECG are listed in table below:

| Parameter (unit) | Criterion value |
|---------------------|-----------------|
| Heart Rate (bpm) | >120 |
| | <50 |
| PR Interval (msec) | ≥ 210 |
| RR Interval (msec) | > 1200 |
| | < 500 |
| QRS Interval (msec) | ≥ 120 |
| | ≤ 50 |
| QT Interval (msec) | ≥ 500 |
| | ≤ 300 |
| QTcF (msec) | > 450 |

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005



| > 480 |
|---------------------------------------|
| > 500 |
| ≤ 300 |
| Increase from baseline > 30 |
| Increase from baseline > 60 |
| Decrease from baseline > 30 |
| Decrease from baseline > 60 |
| > 450 and increase from baseline > 30 |
| > 500 and increase from baseline > 60 |

## 17.6. VITAL SIGNS

The following Vital Signs measurements performed within 37 days after the date of last dose of study medication will be reported for this study:

- Heart rate (bpm)
- Respiratory rate (bpm)
- Body Temperature (C)
- Weight (kg)
- Systolic blood pressure (mmHg)
- Diastolic blood pressure (mmHg)

The following summaries will be provided for vital signs data:

- Observed and change from baseline by visit
- The frequency and percentage of patients with any potentially clinically significant findings defined in section 17.6.2 during the treatment period will be presented.

Listing of vital sign data will also be generated.

#### 17.6.1. VITAL SIGNS SPECIFIC DERIVATIONS

There will be no specific derivations for vital signs.

#### 17.6.2. VITAL SIGNS MARKEDLY ABNORMAL CRITERIA

Markedly abnormal quantitative Vital Signs measurements will be identified and classified in accordance with the following predefined criteria:

| Vital Sign Parameter | Criterion value |
|----------------------|------------------------------------------|
| SBP (mmHg), | Increase from baseline of $> 0 - \le 20$ |
| DBP (mmHg), | $> 20 - \le 40$ |
| Heart rate (bpm) | > 40 |



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



| Vital Sign Parameter | Criterion value |
|----------------------|--------------------------------------|
| | Decrease from baseline of |
| | > 0 - ≤ 20 |
| | > 20 - ≤ 40 |
| | > 40 |
| | Percentage decrease from baseline of |
| | < 5% |
| | $\geq 5 - < 10\%$ |
| | ≥ 10 - < 20% |
| Weight (kg) | ≥ 20% |
| weight (kg) | Percentage increase from baseline of |
| | < 5% |
| | $\geq 5 - < 10\%$ |
| | ≥ 10 - < 20% |
| | $\geq 20\%$ |

## 17.7. PHYSICAL EXAMINATION

The physical examination results collected will be listed.

### 17.8. OTHER SAFETY ASSESSMENTS

#### 17.8.1. ECOG PERFORMANCE STATUS

Summary of ECOG performance status by scheduled visit and change to worst post-baseline value will also be presented. All the ECOG performance status data will also be listed.

#### 17.8.2. ECHOCARDIOGRAM

Baseline and change from baseline on left ventricular ejection fraction (LVEF) will be summarized by dose cohort (only in dose escalation phase) or tumor specific cohorts (only in dose expansion phase) and visit. Also, shift from baseline to worst post-baseline overall evaluation (i.e., normal, abnormal but NCS, abnormal and CS) will be summarized. Individual data will also be listed.

#### 17.8.3. PREGNANCY TEST

Individual pregnancy information will be listed for the SAS.

#### 17.8.4. TUMOR MARKER

CA125 level for patients with ovarian cancer, PSA for patients with prostate cancer, or other tumor markers (as appropriate) should be obtained as clinically indicated or with each tumor assessment. The individual tumor marker test results will be listed for SAS.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

 Effective Date:
 02Dec2019

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.


#### 17.8.5. IMPACT OF COVID-19

The study is conducted during the COVID-19 pandemic, additional data is collected for evaluating the impact of COVID-19. To eliminate potential hazards to patients and study staff due to the COVID-19 pandemic while ensuring patients safety and maintaining data integrity, patients are allowed remote visits during the pandemic. Data listing will be provided.

## 18. REFERENCES

Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). Eur J Cancer. 2009; 45:228-247.

Brookmeyer R., and Crowley J. (1982). A confidence interval for the median survival time. Biometrics, 29-41.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005

## **APPENDIX 1. SCHEDULE OF EVENTS**

Schedule of events is shown as below.

Appendix A Study Schedule of Events

| | | | | | | Treatm | ent² | | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Date<br>Procedure | | | | | | | | | Cycle 4<br>and | Treatment | |
| Frocedure | Scre | ening | | Cv | cle 1 | | Cycl | e 2-3 | onwards | Completion <sup>3</sup> | Follow-up |
| | Day -28<br>to Day - | Day -7<br>to Day - | | Day 8 | Day 15 | Day<br>22 | Day 1 | Day<br>15 | Day 1 of<br>each<br>subsequent<br>cycle (±3d) | 30 (±7) days<br>after permanent<br>treatment | Every 12 (±2) weeks<br>from Treatment |
| Informed consent <sup>1</sup> | 1<br>X | 1 | Day 1 | (±1d) | (±1d) | (±1d) | (±3d) | (±3d) | | discontinuation | Completion Visit |
| Tumor assessment | Λ | | | | | | | | | | |
| (Dose Escalation,<br>Expansion Cohorts<br>C, D, E) | x | | Screen | ning, ther | every 8 ( | ±1) week<br>C7D1, 6 | | ter ( eg C | 3D1, C5D1, | X <sup>4</sup> | |
| Tumor assessment (Dose Expansion Cohorts A and B only) | x | | Screen | ing, C2D | | | d every 8<br>C10D1, | | eks thereafter | X <sup>4</sup> | |
| Medical history,<br>demographics | x | | | | | | | | | | |
| Concomitant<br>medication <sup>5</sup> | Х | Х | х | X | X | X | X | X | х | X | |
| ECOG performance status | | x | X | | X | | X | X | X | X | |
| Vital signs <sup>6</sup> | | X | X | X | X | X | X | X | X | X | |
| Complete physical examination <sup>7</sup> | | X | | | | | | | | | |
| Limited physical<br>examination <sup>7</sup> | | | x | X | X | X | X | X | x | X | |
| Height | X | | | | | | | | | | |
| Hematology <sup>8</sup> Coagulation assay | 1 | X | | X | X | X | X | X | X | X | |
| (aPTT, INR) | | X | | X | X | X | X | X | X | X | |
| Chemistry panel <sup>9</sup> | | X | | X | X | X | X | X | X | X | |
| Urinalysis <sup>10</sup><br>Echocardiogram <sup>11</sup> | X | X | | X (Fye | ry 12 weel | X | X<br>ok after t | he first d | X (asa) | X | |
| Thyroid function<br>test <sup>12</sup> | X | | | A (Eve | ly 12 wee | X3 ± 1 W | X | ne mst d | x | X | |
| Serum pregnancy<br>tests 13 | | х | | | | | | | | X | |
| Urine pregnancy<br>tests <sup>13</sup> | | | | | | | х | | x | | |
| Specific tumor<br>markers <sup>14</sup><br>Dose Escalation,<br>Expansion Cohorts<br>C, D, E) | x | | Scre | eening, th | en every 8 | (±1) we<br>C7D1, | | after: C31 | D1, C5D1, | | |
| Specific tumor<br>markers <sup>14</sup><br>Dose Expansion<br>Cohorts A and B<br>only) | | | Screen | ing, C2D | 1, C3D1 ( | C4D1, an | d every 8 | (±1) wee | eks thereafter | | |
| 12-lead<br>electrocardiogram <sup>15</sup> | | х | х | | х | | х | | x | X | |
| PK plasma sampling | | | | | | | | | 1 15 of Cycle<br>pendix D for | | |
| | | | | | sp | ecific tin | | | • | | |
| Adverse event <sup>16</sup> | X | X | X | X | X | X | X | X | X | X | |
| Fruquintinib<br>treatment | | | Once daily, 3 weeks on/ 1 week off | | | | | | | | |
| Survival follow up <sup>17</sup> | | | | | | | | | | | X |

| Document: | |
|---------------|------------------------|
| Template No.: | Reference: CS WI BS005 |




#### Note:

- A written informed consent form should be obtained prior to any protocol-specific procedure or test. Tests completed within 28
  days prior to enrollment can be used for screening and do not need to be repeated (except hematology, coagulation test, clinical
  chemistry, or urinalysis results).
- Unless otherwise indicated, the visit window during the treatment period will be ± 3 days (± 1 day during cycle 1).
- 3. Patients who complete or prematurely discontinue the study need to return to the study site for a follow-up at 30 (±7) days after the decision to discontinue treatment permanently. Ongoing AEs will be followed until the event has resolved to baseline grade, the event is assessed as stable by the investigator, new anti-tumor treatment is initiated, the patient is lost to follow-up, the patient withdraws consent, or when it has been determined that the study treatment or participation is not the cause of the AE.
- 4. The treatment completion visit tumor assessment can be omitted if treatment ended because of disease progression or the patient had a tumor assessment within 14 days prior to the last dose of study drug.
- Concomitant medication includes any prescribed or over-the-counter medicines. All medication used by patients within 7 days before screening and 30 days after study treatment completion should be recorded. At each visit, all medication used since the prior visit should be recorded.
- Vital signs include blood pressure, heart rate, respiratory rate, and temperature. For patient with a baseline history of
  antihypertensive medications, blood pressure should be monitored at 3 hours (±2 hours) after the daily doses of anti-hypertensive
  medication.
- 7. Please refer to Section 6.3.2 for the assessments that should be completed as part of the Complete and Limited Physical Exams.
- Hematology consists of complete blood count, including red blood cell count, hemoglobin, hematocrit, reticulocyte count, white blood cell count with differential (neutrophils, bands, lymphocytes, eosinophils, monocytes, basophils, and other cells), and platelet count.
- The chemistry panel includes blood urea nitrogen, creatinine and creatinine clearance, sodium, potassium, chlorine, bicarbonate, calcium, magnesium, phosphorus, glucose, alanine aminotransferase, bilirubin (total), aspartate aminotransferase, alkaline phosphatase, lactate dehydrogenase, total cholesterol, triglycerides, uric acid, protein (total) and albumin.
- 10. Urinalysis includes pH, glucose, protein, and blood. A 24-hour urine should be collected from all patients with >1+ proteinuria for quantitative test of urine protein during the screening. If protein ≥2+ during the period of study treatment, a 24-hour urine test should be conducted within 1 week.
- 11. MUGAs are permitted if echocardiograms cannot be performed.
- 12. Includes free T3, free T4, and thyroid-stimulating hormone (TSH).
- 13. Women of childbearing potential will receive a serum pregnancy test during screening and within 30 days after treatment completion, and a urine pregnancy test on Day 1 of each 28-day cycle beginning at Cycle 2. If pregnancy is suspected, additional tests should be completed. In the case of menopausal women, the date of menopause onset should be recorded.
- 14. CA125 level for patients with ovarian cancer, PSA for patients with prostate cancer, or other tumor markers (as appropriate) should be obtained as clinically indicated or with each tumor assessment.
- 15. On Days 1 and 15 in Cycle 1, ECG should be performed at pre-dose and at 3 hours (± 15 minutes) post-dose (around C<sub>max</sub> after single dose and at steady state in order to evaluate concentration-QT relationship for fruquintinib). Untimed ECG will be conducted on Day 1 of each cycle from Cycle 2 and onward.
- 16. After informed consent, all SAEs and concomitant medications will be collected. After initiation of study drug, all AEs and SAEs will be collected until 30 days following the last dose of study drug or a new treatment of anti-tumor therapy, whichever is earlier. After this period, investigators should report only SAEs that are considered to be related to the study drug.
- 17. For subjects in Expansion Cohorts B, C, D, and E Survival follow-up (by telephone) should be performed every 12 (±2) weeks from the date of the Treatment Completion visit. All subsequent anti-tumor therapy and information about ongoing or unresolved study drug-related SAEs will be collected. For the patients that discontinue the study without PD, all available tumor assessment results during survival follow-up will be recorded in the CRF until confirmation of PD. The date and cause of death should be recorded, if applicable. Patients who withdraw consent are encouraged to be followed for survival. If the patient has clearly expressed his/her refusal to be followed after withdrawal of consent, he/she will terminate the study and no survival follow-up will be performed.

| Document: | | |
|-------------|-----|------------------------|
| Template No | D.: | Reference: CS_WI_BS005 |

## APPENDIX 2. PROGRAMMING CONVENTIONS FOR OUTPUTS

#### **Output Conventions**

For more details please refer to the general rules listed in the shell.

#### **Dates & Times**

Depending on data available, dates and times will take the form ddmmyyyyThh:mm:ss.

#### **Spelling Format**

English US.

#### **Presentation of Treatment Groups**

For outputs, treatment groups will be represented as follows and in that order:

| Treatment Group | For Tables |
|---|---|
| Dose Escalation Phase: 3mg QD | Dose Escalation Phase: Fruquintinib 3mg QD |
| Dose Escalation Phase: 5mg QD | Dose Escalation Phase: Fruquintinib 5mg QD |
| Dose Expansion Phase (5mg QD): Cohort A | Dose Expansion Phase: Cohort A |
| Dose Escalation Phase: 5mg QD | Dose Expansion Phase: Dose Escalation |
| + Dose Expansion Phase (5mg QD): Cohort A | Fruquintinib 5mg QD + Cohort A |
| Dose Escalation Phase + Dose Expansion Phase | Dose Expansion Phase: Dose Escalation Phase + |
| | Dose Expansion Phase |
| | (Only for Patient Disposition, Demographic and |
| | Baseline Characteristics, Baseline Cancer |
| | Characteristics tables) |

| Treatment Group | For Listings |
|---|---|
| Dose Escalation Phase: 3mg QD | Dose Escalation Phase: Fruquintinib 3mg QD |
| Dose Escalation Phase: 5mg QD | Dose Escalation Phase: Fruquintinib 5mg QD |
| Dose Expansion Phase (5mg QD): Cohort A | Dose Expansion Phase: Cohort A |

| Treatment Group | For Figures |
|-------------------------------|--------------------------------------------|
| Dose Escalation Phase: 3mg QD | Dose Escalation Phase: Fruquintinib 3mg QD |
| Dose Escalation Phase: 5mg QD | Dose Escalation Phase: Fruquintinib 5mg QD |

Document:


Template No.: Reference: CS\_WI\_BS005




| Treatment Group | For Figures |
|---|---|
| Dose Expansion Phase (5mg QD): Cohort A | Dose Expansion Phase: Cohort A |
| Dose Escalation Phase: 5mg QD | Pooling Dose Escalation 5 mg and Cohort A |
| and Dose Expansion Phase (5mg QD): Cohort A | |
| Dose Escalation Phase: 3mg QD | Dose Escalation 3mg and Pooling Dose |
| + Dose Escalation Phase: 5mg QD | Escalation 5mg and Cohort A |
| and Dose Expansion Phase (5mg QD): Cohort A | |

#### **Presentation of Visits**

For outputs, visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|---------------------|------------|
| Baseline | Baseline |
| Cycle 1 Day 1 | C1D1 |
| Cycle 1 Day 8 | C1D8 |
| Cycle 1 Day 15 | C1D15 |
| Cycle 1 Day 22 | C1D22 |
| Cycle 2 Day 1 | C2D1 |
| Cycle 2 Day 15 | C2D15 |
| Cycle 3 Day 1 | C3D15 |
| Cycle 4 Day 1 | C4D1 |
| Cycle X Day 1 | CXD1 |
| End of Treatment | EOT |

#### **Listings**

All listings will be ordered by the following (unless otherwise indicated in the template):

Assigned treatment group, unless otherwise specified

Center-Patient Number

Date (where applicable)

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005



# APPENDIX 3. BEST OVERALL RESPONSE WHEN CONFIRMATION OF CR AND PR ARE REQUIRED

| | | Best overall | Best Overall Response for |
|---|---|---|---|
| First TPR | Second TPR[a] | response*^ for ORR | ORRUNCONFIRMED |
| CR | CR | CR | CR |
| CR | PR | SD [b] or PD | Unconfirmed CR |
| CR | SD | SD [b] or PD | Unconfirmed CR |
| CR | PD | SD [b] or PD | Unconfirmed CR |
| CR | NE or NA | SD [c] or NE or NA | Unconfirmed CR |
| PR | CR | PR | Unconfirmed CR |
| PR | PR | PR | PR |
| PR | SD | SD [d] | Unconfirmed PR |
| PR | PD | SD [b] or PD | Unconfirmed PR |
| PR | NE or NA | SD [c] or NE or NA | Unconfirmed PR |
| NE | NE | NE | NE |
| NE | CR | SD | Unconfirmed CR |
| NE | PR | SD | Unconfirmed PR |
| NE | SD | SD | SD |
| NE or NA | PD | PD | PD |
| SD | PD | SD [b] or PD | SD [b] or PD |
| SD | CR | SD | SD |
| SD | PR | SD | SD |
| SD | SD | SD | SD |
| SD | NE or NA | SD [c] or NE or NA | SD [c] or NE |
| PD | No further | | |
| | evaluation | PD | PD D. |

CR = Complete Response; NE = Not Evaluable; NA = Not Available; ORR = Objective Response Rate; PD = Progressive Disease; PR= Partial Response; SD = Stable Disease.

[a] The minimum interval for confirmation of CR and PR is 4 weeks.

[b]Best response will be SD if the first time point overall response is after 49 days on study. Otherwise, the best response will be PD.

[c]Best response will be SD if the first time point overall response after 49 days on study. Otherwise, the best response will be NE.

| Document: | |
|---------------------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |
| Effective Date: 02Dec2019 | |

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




[d]Best response will be SD provided the criteria for PD have not been met from the first to second assessment.

- \* A best overall response of SD can only be made after the subject is on study for a minimum of 49 days (counted from Cycle 1 Day 1). If the subject is on study for less than 49 days, any tumor assessment indicating stable disease before this time period will have a best response of NE unless PD is identified.
- ^ Subsequent documentation of a CR may provide confirmation of a previously identified CR even with an intervening NE (e.g., CR NE CR). Subsequent documentation of a PR may provide confirmation of a previously identified PR even with an intervening NE or SD (e.g., PR NE PR or PR SD PR). However, only one (1) intervening NE or SD will be allowed between PRs for confirmation. Note: in the following scenario, PR SD NE PR, the second PR is not a confirmation of the first PR.

 Document:
 2.5

 Author:
 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005



Statistical Analysis Plan 

## APPENDIX 4. VISIT-WINDOW MAPPING

Document:
Author:


Template No.: Reference: CS\_WI\_BS005



Statistical Analysis Plan 

| | Cycle 1 | | Cycle 2-3 | | Cycle 4 and onwards | Post-treatment | | |
|---|---|---|---|---|---|---|---|---|
| Visit | C1D1 | C1D8 | C1D15 | C1D22 | CxD1 | CxD15 | CxD1 | |
| Scheduled Day [a] | 1 | 8 | 15 | 22 | 1 | 15 | 1 | |
| ECOG | Day 1 | | 2 to EOC-3 | | Day -3 to 3 | 4 to EOC-3 | Day -3 to 3 | |
| Vital Sign | Day 1 | 2 to 11 | 12 to 18 | 19 to EOC-3 | Day -3 to 3 | 4 to EOC-3 | Day -3 to 3 | |
| Hematology | | 1 to 11 | 12 to 18 | 19 to EOC-3 | Day -3 to 3 | 4 to EOC-3 | Day -3 to 3 | |
| Coagulation | | 1 to 11 | 12 to 18 | 19 to EOC-3 | Day -3 to 3 | 4 to EOC-3 | Day -3 to 3 | Last dose date of last cycle +8 |
| Clinical Chemistry | | 1 to 11 | 12 to 18 | 19 to EOC-3 | Day -3 to 3 | 4 to EOC-3 | Day -3 to 3 | to last dose date +37 |
| Urinalysis | | 1 to 11 | 12 to 18 | 19 to EOC-3 | Day -3 to 3 | 4 to EOC-3 | Day -3 to 3 | |
| Thyroid function | | 1 to 11 | 12 to 18 | 19 to EOC-3 | Day -3 to 3 | 4 to EOC-3 | Day -3 to 3 | |
| 12-Led ECG | Day 1 | | 2 to EOC-3 | | Day -3 to 3 | | Day -3 to 3 | |

[a] The scheduled day is relative to the Day 1 of each cycle.

Note: The end date of a cycle (EOC) is defined as the one day earlier than the date of Day 1 study drug administration of its next cycle. For the last cycle (where no subsequent cycle if given), the end of cycle will be defined as Day 7 relative to the last dose of the cycle.

#### Tumor Assessment

| I dilloi A33C33iliCiliC | | | | | | |
|---|---|---|---|---|---|---|
| | Cycle 2 | Cycle 3 | Cycle 4 | 8 Weeks after D1 of Cycle 4 | 8 * (X + 1) Weeks after D1 of Cycle 4 [b] | Post-treatment |
| Visit | C2D1 | C3D1 | C4D1 | 8 Weeks after D1 of Cycle 4 | 8 * (X + 1) Weeks after D1 of Cycle 4 [b] | |
| Scheduled Day [a] | 1 | 1 | 1 | 57 | 1 + 7*8 * (X + 1) | |
| Tumor Assessment<br>(Cohort A and B) | -3 to (EOC-3) | -3 to (EOC-3) | -3 to (EOC-3) | End of Cycle 4 to 85 | 28 * (2X + 1) + 2<br>to 28 * (2X + 3) + 1 [d] | |
| | Week 8 | Week 8 * (X + 1) | | | | |
| Visit | Week 8 | Week 8 * (X + 1) [b] | | | | Last dose date of last cycle +8<br>to last dose date +37 |
| Scheduled Day [c] | 57 | 1 + 7*8 * (X + 1) | | | | to last dose date +37 |
| Tumor Assessment<br>(Cohort C, D, and E) | Day 2 to 85 | 28 * (2X + 1) + 2<br>to 28 * (2X + 3) + 1 [d] | | | | |

[a] The scheduled day is relative to the Day 1 for Cycle 2 to Cycle 4, but the subsequent scheduled day is relative to Day 1 of Cycle 4.

Note: The end date of a cycle (EOC) is defined as the one day earlier than the date of Day 1 study drug administration of its next cycle. For the last cycle (where no subsequent cycle if given), the end of cycle will be defined as Day 7 relative to the last dose of the cycle.

| Document: | |
|---------------|------------------------|
| Template No.: | Reference: CS WI BS005 |

Effective Date: 02Dec2019

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

<sup>[</sup>b] X is an intergern starting from 1, and will take maximum value at date of last study drug administration.

<sup>[</sup>c] Scheduled day is relative to Day 1 of Cycle 1.

<sup>[</sup>d] The last windowed visit end by the last dose date.



Statistical Analysis Plan 

#### Echocardiogram

| | | Week 12 * (X + 1) | Post-treatment |
|---|---|---|---|
| Visit | Week 12 | Week 12 * (X + 1) [b] | |
| Scheduled Day [c] | 85 | 1 + 7*12 * (X + 1) | |
| Echocardiogram | Day 2 to 127 | 42 * (2X + 1) + 2<br>to 42 * (2X + 3) + 1 [c] | Last dose date of last cycle +8<br>to last dose date +37 |

<sup>[</sup>a] The scheduled day is relative to the Day 1 of Cycle 1.

| Document: | |
|---------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |

<sup>[</sup>b] X is an intergern starting from 1, and will take maximum value at date of last study drug administration.

<sup>[</sup>c] The last windowed visit end by the last dose date.



Statistical Analysis Plan 

# APPENDIX 5. MEDDRA (VERSION 24.1) PREFERRED TERM LIST FOR AESI CATEGORIES

| AESI Category: Thyroid Dysfunction | | |
|---|---|---|
| Anti-thyroid antibody | Marine Lenhart syndrome | Thyroid size decreased |
| Anti-thyroid antibody decreased | Multifocal fibrosclerosis | Thyroid stimulating hormone deficiency |
| Anti-thyroid antibody increased | Myxoedema | Thyroid stimulating immunoglobulin increased |
| Anti-thyroid antibody positive | Myxoedema coma | Thyroid therapy |
| Antithyroid arthritis syndrome | Orbital decompression | Thyroid tuberculosis |
| Atrophic thyroiditis | Photon radiation therapy to thyroid | Thyroidectomy |
| Autoimmune hypothyroidism | Polyglandular autoimmune syndrome type II | Thyroiditis |
| Autoimmune thyroid disorder | Polyglandular autoimmune syndrome type III | Thyroiditis acute |
| Autoimmune thyroiditis | Post procedural hypothyroidism | Thyroiditis chronic |
| Basedow's disease | Primary hyperthyroidism | Thyroiditis fibrous chronic |
| Biopsy thyroid gland abnormal | Primary hypothyroidism | Thyroiditis subacute |
| Blood thyroid stimulating hormone abnormal | Protein bound iodine decreased | Thyrotoxic cardiomyopathy |
| Blood thyroid stimulating hormone decreased | Protein bound iodine increased | Thyrotoxic crisis |
| Blood thyroid stimulating hormone increased | Radioactive iodine therapy | Thyrotoxic myopathy |
| Butanol-extractable iodine decreased | Radiotherapy to thyroid | Thyrotoxic periodic paralysis |
| Butanol-extractable iodine increased | Reverse tri-iodothyronine decreased | Thyroxin binding globulin abnormal |
| Congenital hypothyroidism | Reverse tri-iodothyronine increased | Thyroxin binding globulin decreased |
| Congenital thyroid disorder | Secondary hyperthyroidism | Thyroxin binding globulin increased |
| Endocrine ophthalmopathy | Secondary hypothyroidism | Thyroxine abnormal |
| Euthyroid sick syndrome | Silent thyroiditis | Thyroxine decreased |
| Exophthalmos | Tertiary hypothyroidism | Thyroxine free abnormal |
| Free thyroxine index abnormal | Thyreostatic therapy | Thyroxine free decreased |
| Free thyroxine index decreased | Thyroglobulin absent | Thyroxine free increased |
| Free thyroxine index increased | Thyroglobulin decreased | Thyroxine increased |
| Gamma radiation therapy to thyroid | Thyroglobulin increased | Thyroxine therapy |

| Document: |
|-----------|

Template No.: Reference: CS\_WI\_BS005



Statistical Analysis Plan 

| Generalised resistance to thyroid hormone | Thyroglobulin present | Toxic goitre |
|---|---|---|
| Goitre | Thyroid atrophy | Toxic nodular goitre |
| Hashimoto's encephalopathy | Thyroid autotransplantation | Transient hypothyroxinaemia of prematurity |
| Hashitoxicosis | Thyroid dermatopathy | Tri-iodothyronine abnormal |
| Hyperthyroidism | Thyroid disorder | Tri-iodothyronine decreased |
| Hypothyroidic goitre | Thyroid dysfunction in pregnancy | Tri-iodothyronine free abnormal |
| Hypothyroidism | Thyroid electron radiation therapy | Tri-iodothyronine free decreased |
| Immune-mediated hyperthyroidism | Thyroid function test abnormal | Tri-iodothyronine free increased |
| Immune-mediated hypothyroidism | Thyroid gland scan abnormal | Tri-iodothyronine free normal |
| Immune-mediated thyroiditis | Thyroid hemiagenesis | Tri-iodothyronine increased |
| Inappropriate thyroid stimulating hormone secretion | Thyroid hormone replacement therapy | Tri-iodothyronine uptake abnormal |
| Infectious thyroiditis | Thyroid hormones decreased | Tri-iodothyronine uptake decreased |
| Iodine uptake abnormal | Thyroid hormones increased | Tri-iodothyronine uptake increased |
| Iodine uptake decreased | Thyroid operation | Ultrasound thyroid abnormal |
| Iodine uptake increased | Thyroid pain | X-ray therapy to thyroid |
| Malignant exophthalmos | Thyroid releasing hormone challenge test abnormal | |
| | AESI Category: Proteinuria | |
| Albumin globulin ratio increased | Beta 2 microglobulin urine increased | Protein urine |
| Albumin urine present | Globulinuria | Protein urine present |
| Albuminuria | Microalbuminuria | Proteinuria |
| Bence Jones protein urine present | Myoglobinuria | Urine albumin/creatinine ratio increased |
| Bence Jones proteinuria | Orthostatic proteinuria | Urine protein/creatinine ratio abnormal |
| | | Urine protein/creatinine ratio increased |
| | AESI Category: Hypertension | |
| Accelerated hypertension | Eclampsia | Metabolic syndrome |
| Aldosterone urine abnormal | Ectopic aldosterone secretion | Metanephrine urine abnormal |
| Aldosterone urine increased | Ectopic renin secretion | Metanephrine urine increased |

 Document:
 Author:
 2.5

 18Feb2022

 Template No.:
 Reference: CS\_WI\_BS005



## Statistical Analysis Plan 

| Angiotensin converting enzyme increased | Endocrine hypertension | Neurogenic hypertension |
|---|---|---|
| Angiotensin I increased | Epinephrine abnormal | Non-dipping |
| Angiotensin II increased | Epinephrine increased | Norepinephrine abnormal |
| Angiotensin II receptor type 1 antibody positive | Essential hypertension | Norepinephrine increased |
| Blood aldosterone abnormal | Gestational hypertension | Normetanephrine urine increased |
| Blood aldosterone increased | HELLP syndrome | Orthostatic hypertension |
| Blood catecholamines abnormal | Hyperaldosteronism | Page kidney |
| Blood catecholamines increased | Hypertension | Postoperative hypertension |
| Blood pressure abnormal | Hypertension neonatal | Pre-eclampsia |
| Blood pressure ambulatory abnormal | Hypertensive angiopathy | Prehypertension |
| Blood pressure ambulatory increased | Hypertensive cardiomegaly | Procedural hypertension |
| Blood pressure diastolic abnormal | Hypertensive cardiomyopathy | Pseudoaldosteronism |
| Blood pressure diastolic increased | Hypertensive cerebrovascular disease | Renal hypertension |
| Blood pressure fluctuation | Hypertensive crisis | Renal sympathetic nerve ablation |
| Blood pressure inadequately controlled | Hypertensive emergency | Renal vascular resistance increased |
| Blood pressure increased | Hypertensive encephalopathy | Renin abnormal |
| Blood pressure management | Hypertensive end-organ damage | Renin increased |
| Blood pressure orthostatic abnormal | Hypertensive heart disease | Renin-angiotensin system inhibition |
| Blood pressure orthostatic increased | Hypertensive nephropathy | Renovascular hypertension |
| Blood pressure systolic abnormal | Hypertensive urgency | Retinopathy hypertensive |
| Blood pressure systolic increased | Labile blood pressure | Secondary aldosteronism |
| Catecholamine crisis | Labile hypertension | Secondary hypertension |
| Catecholamines urine abnormal | Malignant hypertension | Superimposed pre-eclampsia |
| Catecholamines urine increased | Malignant hypertensive heart disease | Supine hypertension |
| Dialysis induced hypertension | Malignant renal hypertension | Systolic hypertension |
| Diastolic hypertension | Maternal hypertension affecting foetus | Tyramine reaction |
| Diuretic therapy | Mean arterial pressure increased | Withdrawal hypertension |
| | AESI Category: Haemorrhages | |

 Document:
 2.5

 Author:
 18Feb2022

Template No.: Reference: CS\_WI\_BS005



## Statistical Analysis Plan 

| Abdominal wall haematoma | Haemophilic pseudotumour | Petechiae |
|---|---|---|
| Abdominal wall haemorrhage | Haemoptysis | Pharyngeal contusion |
| Abnormal uterine bleeding | Haemorrhage | Pharyngeal haematoma |
| Abnormal withdrawal bleeding | Haemorrhage coronary artery | Pharyngeal haemorrhage |
| Achenbach syndrome | Haemorrhage foetal | Pituitary apoplexy |
| Acute haemorrhagic leukoencephalitis | Haemorrhage in pregnancy | Pituitary haemorrhage |
| Acute haemorrhagic ulcerative colitis | Haemorrhage intracranial | Placenta praevia haemorrhage |
| Administration site bruise | Haemorrhage neonatal | Polymenorrhagia |
| Administration site haematoma | Haemorrhage subcutaneous | Post abortion haemorrhage |
| Administration site haemorrhage | Haemorrhage subepidermal | Post procedural contusion |
| Adrenal haematoma | Haemorrhage urinary tract | Post procedural haematoma |
| Adrenal haemorrhage | Haemorrhagic adrenal infarction | Post procedural haematuria |
| Anal fissure haemorrhage | Haemorrhagic arteriovenous malformation | Post procedural haemorrhage |
| Anal haemorrhage | Haemorrhagic ascites | Post transfusion purpura |
| Anal ulcer haemorrhage | Haemorrhagic breast cyst | Postmenopausal haemorrhage |
| Anastomotic haemorrhage | Haemorrhagic cerebellar infarction | Postpartum haemorrhage |
| Anastomotic ulcer haemorrhage | Haemorrhagic cerebral infarction | Post-traumatic punctate intraepidermal haemorrhage |
| Aneurysm ruptured | Haemorrhagic cyst | Premature separation of placenta |
| Angina bullosa haemorrhagica | Haemorrhagic diathesis | Procedural haemorrhage |
| Anorectal varices haemorrhage | Haemorrhagic disease of newborn | Proctitis haemorrhagic |
| Anticoagulant-related nephropathy | Haemorrhagic disorder | Prostatic haemorrhage |
| Antiplatelet reversal therapy | Haemorrhagic erosive gastritis | Pulmonary alveolar haemorrhage |
| Aortic aneurysm rupture | Haemorrhagic gastroenteritis | Pulmonary contusion |
| Aortic dissection rupture | Haemorrhagic hepatic cyst | Pulmonary haematoma |
| Aortic intramural haematoma | Haemorrhagic infarction | Pulmonary haemorrhage |
| Aortic perforation | Haemorrhagic necrotic pancreatitis | Pulmonary haemorrhage neonatal |
| Aortic rupture | Haemorrhagic occlusive retinal vasculitis | Puncture site bruise |
| Aponeurosis contusion | Haemorrhagic ovarian cyst | Puncture site haematoma |
| Application site bruise | Haemorrhagic stroke | Puncture site haemorrhage |

Document:
Author:


Reference: CS\_WI\_BS005

Effective Date: 02Dec2019

Template No.:



## Statistical Analysis Plan 

| Application site haematoma | Haemorrhagic thyroid cyst | Purpura |
|---|---|---|
| Application site haemorrhage | Haemorrhagic transformation stroke | Purpura fulminans |
| Application site purpura | Haemorrhagic tumour necrosis | Purpura neonatal |
| Arterial haemorrhage | Haemorrhagic urticaria | Purpura non-thrombocytopenic |
| Arterial intramural haematoma | Haemorrhagic vasculitis | Purpura senile |
| Arterial perforation | Haemorrhoidal haemorrhage | Putamen haemorrhage |
| Arterial rupture | Haemostasis | Radiation associated haemorrhage |
| Arteriovenous fistula site haematoma | Haemothorax | Rectal haemorrhage |
| Arteriovenous fistula site haemorrhage | Heavy menstrual bleeding | Rectal ulcer haemorrhage |
| Arteriovenous graft site haematoma | Henoch-Schonlein purpura | Renal artery perforation |
| Arteriovenous graft site haemorrhage | Hepatic haemangioma rupture | Renal cyst haemorrhage |
| Astringent therapy | Hepatic haematoma | Renal haematoma |
| Atrial rupture | Hepatic haemorrhage | Renal haemorrhage |
| Auricular haematoma | Hereditary haemorrhagic telangiectasia | Respiratory tract haemorrhage |
| Basal ganglia haematoma | Hyperfibrinolysis | Respiratory tract haemorrhage neonatal |
| Basal ganglia haemorrhage | Hypergammaglobulinaemic purpura of Waldenstrom | Retinal aneurysm rupture |
| Basilar artery perforation | Hyphaema | Retinal haemorrhage |
| Bladder tamponade | Iliac artery perforation | Retinopathy haemorrhagic |
| Bleeding varicose vein | Iliac artery rupture | Retroperitoneal haematoma |
| Blood blister | Iliac vein perforation | Retroperitoneal haemorrhage |
| Blood loss anaemia | Immune thrombocytopenia | Retroplacental haematoma |
| Blood urine | Implant site bruising | Ruptured cerebral aneurysm |
| Blood urine present | Implant site haematoma | Scleral haematoma |
| Bloody discharge | Implant site haemorrhage | Scleral haemorrhage |
| Bloody peritoneal effluent | Incision site haematoma | Scrotal haematocoele |
| Bone contusion | Incision site haemorrhage | Scrotal haematoma |
| Bone marrow haemorrhage | Increased tendency to bruise | Scrotal haemorrhage |
| Brain contusion | Induced abortion haemorrhage | Shock haemorrhagic |
| Brain stem haematoma | Inferior vena cava perforation | Skin haemorrhage |

Document:
Author:


Reference: CS\_WI\_BS005

Template No.:



## Statistical Analysis Plan 

| Brain stem haemorrhage | Infusion site bruising | Skin neoplasm bleeding |
|---|---|---|
| Brain stem microhaemorrhage | Infusion site haematoma | Skin ulcer haemorrhage |
| Breast haematoma | Infusion site haemorrhage | Small intestinal haemorrhage |
| Breast haemorrhage | Injection site bruising | Small intestinal ulcer haemorrhage |
| Broad ligament haematoma | Injection site haematoma | Soft tissue haemorrhage |
| Bronchial haemorrhage | Injection site haemorrhage | Spermatic cord haemorrhage |
| Bronchial varices haemorrhage | Instillation site bruise | Spinal cord haematoma |
| Bullous haemorrhagic dermatosis | Instillation site haematoma | Spinal cord haemorrhage |
| Bursal haematoma | Instillation site haemorrhage | Spinal epidural haematoma |
| Cardiac contusion | Intermenstrual bleeding | Spinal epidural haemorrhage |
| Carotid aneurysm rupture | Internal haemorrhage | Spinal subarachnoid haemorrhage |
| Carotid artery perforation | Intestinal haematoma | Spinal subdural haematoma |
| Catheter site bruise | Intestinal haemorrhage | Spinal subdural haemorrhage |
| Catheter site haematoma | Intestinal varices haemorrhage | Spleen contusion |
| Catheter site haemorrhage | Intra-abdominal haematoma | Splenic artery perforation |
| Central nervous system haemorrhage | Intra-abdominal haemorrhage | Splenic haematoma |
| Cephalhaematoma | Intracerebral haematoma evacuation | Splenic haemorrhage |
| Cerebellar haematoma | Intracranial haematoma | Splenic varices haemorrhage |
| Cerebellar haemorrhage | Intracranial tumour haemorrhage | Splinter haemorrhages |
| Cerebellar microhaemorrhage | Intraocular haematoma | Spontaneous haematoma |
| Cerebral aneurysm perforation | Intrapartum haemorrhage | Spontaneous haemorrhage |
| Cerebral aneurysm ruptured syphilitic | Intratumoural haematoma | Stoma site haemorrhage |
| Cerebral arteriovenous malformation haemorrhagic | Intraventricular haemorrhage | Stomatitis haemorrhagic |
| Cerebral artery perforation | Intraventricular haemorrhage neonatal | Subarachnoid haematoma |
| Cerebral cyst haemorrhage | Iris haemorrhage | Subarachnoid haemorrhage |
| Cerebral haematoma | Joint microhaemorrhage | Subarachnoid haemorrhage neonatal |
| Cerebral haemorrhage | Jugular vein haemorrhage | Subcapsular hepatic haematoma |
| Cerebral haemorrhage foetal | Kidney contusion | Subcapsular renal haematoma |
| Cerebral haemorrhage neonatal | Lacrimal haemorrhage | Subcapsular splenic haematoma |

Document:
Author:


2.5

Template No.: Reference: CS\_WI\_BS005



## Statistical Analysis Plan 

| Cerebral microhaemorrhage | Large intestinal haemorrhage | Subchorionic haematoma |
|---|---|---|
| Cervix haematoma uterine | Large intestinal ulcer haemorrhage | Subchorionic haemorrhage |
| Cervix haemorrhage uterine | Laryngeal haematoma | Subclavian artery perforation |
| Chest wall haematoma | Laryngeal haemorrhage | Subclavian vein perforation |
| Choroidal haematoma | Lip haematoma | Subcutaneous haematoma |
| Choroidal haemorrhage | Lip haemorrhage | Subdural haematoma |
| Chronic gastrointestinal bleeding | Liver contusion | Subdural haematoma evacuation |
| Chronic pigmented purpura | Lower gastrointestinal haemorrhage | Subdural haemorrhage |
| Ciliary body haemorrhage | Lower limb artery perforation | Subdural haemorrhage neonatal |
| Coital bleeding | Lymph node haemorrhage | Subendocardial haemorrhage |
| Colonic haematoma | Mallory-Weiss syndrome | Subgaleal haematoma |
| Conjunctival haemorrhage | Mediastinal haematoma | Subgaleal haemorrhage |
| Contusion | Mediastinal haemorrhage | Subretinal haematoma |
| Corneal bleeding | Medical device site bruise | Superior vena cava perforation |
| Cullen's sign | Medical device site haematoma | Testicular haemorrhage |
| Cystitis haemorrhagic | Medical device site haemorrhage | Thalamus haemorrhage |
| Deep dissecting haematoma | Melaena | Third stage postpartum haemorrhage |
| Diarrhoea haemorrhagic | Melaena neonatal | Thoracic haemorrhage |
| Disseminated intravascular coagulation | Meningorrhagia | Thrombocytopenic purpura |
| Diverticulitis intestinal haemorrhagic | Menometrorrhagia | Thrombotic thrombocytopenic purpura |
| Diverticulum intestinal haemorrhagic | Mesenteric haematoma | Thyroid haemorrhage |
| Duodenal ulcer haemorrhage | Mesenteric haemorrhage | Tongue haematoma |
| Duodenitis haemorrhagic | Mouth haemorrhage | Tongue haemorrhage |
| Ear haemorrhage | Mucocutaneous haemorrhage | Tonsillar haemorrhage |
| Ecchymosis | Mucosal haemorrhage | Tooth pulp haemorrhage |
| Encephalitis haemorrhagic | Muscle contusion | Tooth socket haemorrhage |
| Enterocolitis haemorrhagic | Muscle haemorrhage | Tracheal haemorrhage |
| Epidural haemorrhage | Myocardial haemorrhage | Traumatic haematoma |
| Epistaxis | Myocardial rupture | Traumatic haemorrhage |

Document:
Author:


Template No.: Reference: CS\_WI\_BS005

18Feb2022



#### Statistical Analysis Plan 

| Exsanguination | Naevus haemorrhage | Traumatic haemothorax |
|---|---|---|
| Extra-axial haemorrhage | Nail bed bleeding | Traumatic intracranial haematoma |
| Extradural haematoma | Nasal septum haematoma | Traumatic intracranial haemorrhage |
| Extradural haematoma evacuation | Neonatal gastrointestinal haemorrhage | Tumour haemorrhage |
| Extravasation blood | Nephritis haemorrhagic | Ulcer haemorrhage |
| Eye contusion | Nipple exudate bloody | Umbilical cord haemorrhage |
| Eye haematoma | Occult blood positive | Umbilical haematoma |
| Eye haemorrhage | Ocular retrobulbar haemorrhage | Umbilical haemorrhage |
| Eyelid bleeding | Oesophageal haemorrhage | Upper gastrointestinal haemorrhage |
| Eyelid contusion | Oesophageal intramural haematoma | Ureteric haemorrhage |
| Eyelid haematoma | Oesophageal ulcer haemorrhage | Urethral haemorrhage |
| Femoral artery perforation | Oesophageal varices haemorrhage | Urinary bladder haematoma |
| Femoral vein perforation | Oesophagitis haemorrhagic | Urinary bladder haemorrhage |
| Foetal-maternal haemorrhage | Omental haemorrhage | Urinary occult blood |
| Fothergill sign positive | Optic disc haemorrhage | Urinary occult blood positive |
| Gallbladder haematoma | Optic nerve sheath haemorrhage | Urogenital haemorrhage |
| Gastric haemorrhage | Oral blood blister | Uterine haematoma |
| Gastric occult blood positive | Oral contusion | Uterine haemorrhage |
| Gastric ulcer haemorrhage | Oral mucosa haematoma | Vaccination site bruising |
| Gastric ulcer haemorrhage, obstructive | Oral purpura | Vaccination site haematoma |
| Gastric varices haemorrhage | Orbital haematoma | Vaccination site haemorrhage |
| Gastritis alcoholic haemorrhagic | Orbital haemorrhage | Vaginal haematoma |
| Gastritis haemorrhagic | Osteorrhagia | Vaginal haemorrhage |
| Gastroduodenal haemorrhage | Ovarian haematoma | Varicose vein ruptured |
| Gastrointestinal anastomotic haemorrhage | Ovarian haemorrhage | Vascular access site bruising |
| Gastrointestinal haemorrhage | Palpable purpura | Vascular access site haematoma |
| Gastrointestinal polyp haemorrhage | Pancreatic haemorrhage | Vascular access site haemorrhage |
| Gastrointestinal ulcer haemorrhage | Pancreatic pseudocyst haemorrhage | Vascular access site rupture |
| Gastrointestinal vascular malformation haemorrhagic | Pancreatitis haemorrhagic | Vascular anastomotic haemorrhage |

Document: Author: Version Number: Version Date:

Template No.: Reference: CS\_WI\_BS005



Statistical Analysis Plan 

| Genital contusion | Papillary muscle haemorrhage | Vascular graft haemorrhage |
|---|---|---|
| Genital haemorrhage | Paranasal sinus haematoma | Vascular pseudoaneurysm ruptured |
| Gingival bleeding | Paranasal sinus haemorrhage | Vascular purpura |
| Graft haemorrhage | Parathyroid haemorrhage | Vascular rupture |
| Grey Turner's sign | Parotid gland haemorrhage | Vein rupture |
| Haemangioma rupture | Pelvic haematoma | Venous haemorrhage |
| Haemarthrosis | Pelvic haematoma obstetric | Venous perforation |
| Haematemesis | Pelvic haemorrhage | Ventricle rupture |
| Haematochezia | Penile contusion | Vertebral artery perforation |
| Haematocoele | Penile haematoma | Vessel puncture site bruise |
| Haematoma | Penile haemorrhage | Vessel puncture site haematoma |
| Haematoma evacuation | Peptic ulcer haemorrhage | Vessel puncture site haemorrhage |
| Haematoma infection | Pericardial haemorrhage | Vitreous haematoma |
| Haematoma muscle | Perineal haematoma | Vitreous haemorrhage |
| Haematosalpinx | Periorbital haematoma | Vulval haematoma |
| Haematospermia | Periorbital haemorrhage | Vulval haematoma evacuation |
| Haematotympanum | Periosteal haematoma | Vulval haemorrhage |
| Haematuria | Peripartum haemorrhage | Withdrawal bleed |
| Haematuria traumatic | Peripheral artery aneurysm rupture | Wound haematoma |
| Haemobilia | Peripheral artery haematoma | Wound haemorrhage |
| Haemoperitoneum | Peripheral exudative haemorrhagic chorioretinopathy | |
| Haemophilic arthropathy | Peritoneal haematoma | |
| | Periventricular haemorrhage neonatal | |
| | AESI Category: Gastrointestinal perforation | |
| Abdominal abscess | Focal peritonitis | Oesophageal perforation |
| Abdominal hernia perforation | Gastric fistula | Oesophageal rupture |
| Abdominal wall abscess | Gastric fistula repair | Oesophageal ulcer perforation |
| Abscess intestinal | Gastric perforation | Oesophageal-pulmonary fistula |

| Document: |
|-----------|

Template No.: Reference: CS\_WI\_BS005



## Statistical Analysis Plan 

| Acquired tracheo-oesophageal fistula | Gastric ulcer perforation | Oesophagobronchial fistula |
|---|---|---|
| Anal abscess | Gastric ulcer perforation, obstructive | Oesophagomediastinal fistula |
| Anal fistula | Gastrointestinal anastomotic leak | Oesophagopleural fistula |
| Anal fistula infection | Gastrointestinal fistula | Pancreatic fistula |
| Anal fistula repair | Gastrointestinal fistula repair | Pancreatic fistula repair |
| Anastomotic ulcer perforation | Gastrointestinal perforation | Peptic ulcer perforation |
| Anovulvar fistula | Gastrointestinal ulcer perforation | Peptic ulcer perforation, obstructive |
| Aortoenteric fistula | Gastropleural fistula | Peptic ulcer repair |
| Aorto-oesophageal fistula | Gastrosplenic fistula | Perforated ulcer |
| Appendiceal abscess | Ileal perforation | Perineal abscess |
| Appendicitis perforated | Ileal ulcer perforation | Perirectal abscess |
| Arterioenteric fistula | Incisional hernia perforation | Peritoneal abscess |
| Atrio-oesophageal fistula | Inguinal hernia perforation | Peritoneocutaneous fistula |
| Chemical peritonitis | Intestinal fistula | Peritonitis |
| Colon fistula repair | Intestinal fistula infection | Peritonitis bacterial |
| Colonic abscess | Intestinal fistula repair | Pneumoperitoneum |
| Colonic fistula | Intestinal perforation | Pneumoretroperitoneum |
| Colo-urethral fistula | Intestinal ulcer perforation | Procedural intestinal perforation |
| Diverticular fistula | Jejunal perforation | Rectal abscess |
| Diverticular perforation | Jejunal ulcer perforation | Rectal fistula repair |
| Diverticulitis intestinal perforated | Large intestinal ulcer perforation | Rectal perforation |
| Douglas' abscess | Large intestine perforation | Rectoprostatic fistula |
| Duodenal perforation | Lower gastrointestinal perforation | Rectourethral fistula |
| Duodenal rupture | Mesenteric abscess | Retroperitoneal abscess |
| Duodenal ulcer perforation | Neonatal intestinal perforation | Small intestinal perforation |
| Duodenal ulcer perforation, obstructive | Oesophageal abscess | Small intestinal ulcer perforation |
| Duodenal ulcer repair | Oesophageal fistula | Spontaneous bacterial peritonitis |
| Enterocolonic fistula | Oesophageal fistula repair | Umbilical hernia perforation |
| Enterocutaneous fistula | | Upper gastrointestinal perforation |

Document:
Author:


18Feb2022

2.5

Template No.:

Reference: CS\_WI\_BS005

18Feb2022



## Statistical Analysis Plan 

| Fistula of small intestine | | |
|---|---|---|
| | APGIC ( F. L. | |
| | AESI Category: Embolic and thrombotic | |
| Acute aortic syndrome | Embolism venous | Pseudo-occlusion of internal carotid artery |
| Acute myocardial infarction | Endarterectomy | Pulmonary artery occlusion |
| Administration site thrombosis | Eye infarction | Pulmonary artery therapeutic procedure |
| Adrenal thrombosis | Femoral artery embolism | Pulmonary artery thrombosis |
| Amaurosis | Fluorescence angiogram abnormal | Pulmonary embolism |
| Amaurosis fugax | Foetal cerebrovascular disorder | Pulmonary endarterectomy |
| Angiogram abnormal | Foetal vascular malperfusion | Pulmonary infarction |
| Angiogram cerebral abnormal | Gastric infarction | Pulmonary microemboli |
| Angiogram peripheral abnormal | Graft thrombosis | Pulmonary thrombosis |
| Angioplasty | Haemorrhagic adrenal infarction | Pulmonary tumour thrombotic microangiopathy |
| Antiphospholipid syndrome | Haemorrhagic cerebral infarction | Pulmonary vein occlusion |
| Aortic bypass | Haemorrhagic infarction | Pulmonary veno-occlusive disease |
| Aortic embolus | Haemorrhagic stroke | Pulmonary venous thrombosis |
| Aortic surgery | Haemorrhagic transformation stroke | Quadriparesis |
| Aortic thrombosis | Haemorrhoids thrombosed | Quadriplegia |
| Aortogram abnormal | Hemiparesis | Renal artery angioplasty |
| Application site thrombosis | Hemiplegia | Renal artery occlusion |
| Arterectomy | Heparin-induced thrombocytopenia | Renal artery thrombosis |
| Arterectomy with graft replacement | Hepatic artery embolism | Renal embolism |
| Arterial angioplasty | Hepatic artery occlusion | Renal infarct |
| Arterial bypass operation | Hepatic artery thrombosis | Renal vascular thrombosis |
| Arterial graft | Hepatic infarction | Renal vein embolism |
| Arterial occlusive disease | Hepatic vascular thrombosis | Renal vein occlusion |
| Arterial revascularisation | Hepatic vein embolism | Renal vein thrombosis |
| Arterial stent insertion | Hepatic vein occlusion | Renal-limited thrombotic microangiopathy |
| Arterial therapeutic procedure | Hepatic vein thrombosis | Retinal artery embolism |

Document:
Author:

Reference: CS\_WI\_BS005


Template No.:



## Statistical Analysis Plan 

| Arterial thrombosis | Homans' sign positive | Retinal artery occlusion |
|---|---|---|
| Arteriogram abnormal | Hypothenar hammer syndrome | Retinal artery thrombosis |
| Arteriogram carotid abnormal | Iliac artery embolism | Retinal infarction |
| Arteriotomy | Iliac artery occlusion | Retinal vascular thrombosis |
| Arteriovenous fistula occlusion | Iliac vein occlusion | Retinal vein occlusion |
| Arteriovenous fistula thrombosis | Implant site thrombosis | Retinal vein thrombosis |
| Arteriovenous graft thrombosis | Incision site vessel occlusion | Revascularisation procedure |
| Artificial blood vessel occlusion | Infarction | Shunt occlusion |
| Aseptic cavernous sinus thrombosis | Inferior vena cava syndrome | Shunt thrombosis |
| Atherectomy | Inferior vena caval occlusion | SI QIII TIII pattern |
| Atherosclerotic plaque rupture | Infusion site thrombosis | Silent myocardial infarction |
| Atrial appendage closure | Injection site thrombosis | Spinal artery embolism |
| Atrial appendage resection | Inner ear infarction | Spinal artery thrombosis |
| Atrial thrombosis | Instillation site thrombosis | Spinal cord infarction |
| Autoimmune heparin-induced thrombocytopenia | Internal capsule infarction | Spinal stroke |
| Axillary vein thrombosis | Intestinal infarction | Splenic artery thrombosis |
| Basal ganglia infarction | Intra-aortic balloon placement | Splenic embolism |
| Basal ganglia stroke | Intracardiac mass | Splenic infarction |
| Basilar artery occlusion | Intracardiac thrombus | Splenic thrombosis |
| Basilar artery thrombosis | Intraoperative cerebral artery occlusion | Splenic vein occlusion |
| Blindness transient | Ischaemic cerebral infarction | Splenic vein thrombosis |
| Bone infarction | Ischaemic stroke | Stoma site thrombosis |
| Brachiocephalic artery occlusion | Jugular vein embolism | Stress cardiomyopathy |
| Brachiocephalic vein occlusion | Jugular vein occlusion | Stroke in evolution |
| Brachiocephalic vein thrombosis | Jugular vein thrombosis | Strokectomy |
| Brain stem embolism | Lacunar infarction | Subclavian artery embolism |
| Brain stem infarction | Lambl's excrescences | Subclavian artery occlusion |
| Brain stem stroke | Left atrial appendage closure implant | Subclavian artery thrombosis |
| Brain stem thrombosis | Leriche syndrome | Subclavian vein occlusion |

Document:
Author:


Reference: CS\_WI\_BS005

Template No.:



## Statistical Analysis Plan 

| Budd-Chiari syndrome | Mahler sign | Subclavian vein thrombosis |
|---|---|---|
| Capsular warning syndrome | May-Thurner syndrome | Superficial vein thrombosis |
| Cardiac ventricular thrombosis | Medical device site thrombosis | Superior sagittal sinus thrombosis |
| Carotid angioplasty | Mesenteric arterial occlusion | Superior vena cava occlusion |
| Carotid arterial embolus | Mesenteric arteriosclerosis | Superior vena cava syndrome |
| Carotid artery bypass | Mesenteric artery embolism | Surgical vascular shunt |
| Carotid artery occlusion | Mesenteric artery stenosis | Testicular infarction |
| Carotid artery stent insertion | Mesenteric artery stent insertion | Thalamic infarction |
| Carotid artery thrombosis | Mesenteric artery thrombosis | Thrombectomy |
| Carotid endarterectomy | Mesenteric vascular insufficiency | Thromboangiitis obliterans |
| Catheter directed thrombolysis | Mesenteric vascular occlusion | Thromboembolectomy |
| Catheter site thrombosis | Mesenteric vein thrombosis | Thrombolysis |
| Catheterisation venous | Mesenteric venous occlusion | Thrombophlebitis |
| Cavernous sinus thrombosis | Microembolism | Thrombophlebitis migrans |
| Central venous catheterisation | Monoparesis | Thrombophlebitis neonatal |
| Cerebellar artery occlusion | Monoplegia | Thrombosed varicose vein |
| Cerebellar artery thrombosis | Muscle infarction | Thrombosis |
| Cerebellar embolism | Myocardial infarction | Thrombosis corpora cavernosa |
| Cerebellar infarction | Myocardial necrosis | Thrombosis in device |
| Cerebral artery embolism | Obstetrical pulmonary embolism | Thrombosis mesenteric vessel |
| Cerebral artery occlusion | Obstructive shock | Thrombosis prophylaxis |
| Cerebral artery stent insertion | Ophthalmic artery occlusion | Thrombosis with thrombocytopenia syndrome |
| Cerebral artery thrombosis | Ophthalmic artery thrombosis | Thrombotic cerebral infarction |
| Cerebral congestion | Ophthalmic vein thrombosis | Thrombotic microangiopathy |
| Cerebral hypoperfusion | Optic nerve infarction | Thrombotic stroke |
| Cerebral infarction | Ovarian vein thrombosis | Thrombotic thrombocytopenic purpura |
| Cerebral infarction foetal | Paget-Schroetter syndrome | Thyroid infarction |
| Cerebral ischaemia | Pancreatic infarction | Transient ischaemic attack |
| Cerebral microembolism | Papillary muscle infarction | Transverse sinus thrombosis |

Document:
Author:


Reference: CS\_WI\_BS005

Template No.:

18Feb2022



## Statistical Analysis Plan 

| Cerebral microinfarction | Paradoxical embolism | Truncus coeliacus thrombosis |
|---|---|---|
| Cerebral septic infarct | Paraneoplastic thrombosis | Tumour embolism |
| Cerebral thrombosis | Paraparesis | Tumour thrombectomy |
| Cerebral vascular occlusion | Paraplegia | Tumour thrombosis |
| Cerebral venous sinus thrombosis | Paresis | Ultrasonic angiogram abnormal |
| Cerebral venous thrombosis | Pelvic venous thrombosis | Ultrasound Doppler abnormal |
| Cerebrospinal thrombotic tamponade | Penile artery occlusion | Umbilical cord occlusion |
| Cerebrovascular accident | Penile vein thrombosis | Umbilical cord thrombosis |
| Cerebrovascular accident prophylaxis | Percutaneous coronary intervention | Vaccination site thrombosis |
| Cerebrovascular disorder | Peripheral arterial occlusive disease | Vascular access site thrombosis |
| Cerebrovascular insufficiency | Peripheral arterial reocclusion | Vascular device occlusion |
| Cerebrovascular operation | Peripheral artery angioplasty | Vascular graft |
| Cerebrovascular stenosis | Peripheral artery bypass | Vascular graft occlusion |
| Choroidal infarction | Peripheral artery occlusion | Vascular graft thrombosis |
| Coeliac artery occlusion | Peripheral artery stent insertion | Vascular operation |
| Collateral circulation | Peripheral artery surgery | Vascular pseudoaneurysm thrombosis |
| Compression garment application | Peripheral artery thrombosis | Vascular stent insertion |
| Coronary angioplasty | Peripheral embolism | Vascular stent occlusion |
| Coronary arterial stent insertion | Peripheral endarterectomy | Vascular stent thrombosis |
| Coronary artery bypass | Peripheral revascularisation | Vasodilation procedure |
| Coronary artery embolism | Peripheral vein occlusion | Vena cava embolism |
| Coronary artery occlusion | Peripheral vein thrombus extension | Vena cava filter insertion |
| Coronary artery reocclusion | Phlebectomy | Vena cava filter removal |
| Coronary artery surgery | Pituitary infarction | Vena cava thrombosis |
| Coronary artery thrombosis | Placental infarction | Venogram abnormal |
| Coronary bypass thrombosis | Pneumatic compression therapy | Venoocclusive disease |
| Coronary endarterectomy | Popliteal artery entrapment syndrome | Venoocclusive liver disease |
| Coronary revascularisation | Portal shunt procedure | Venous angioplasty |
| Coronary vascular graft occlusion | Portal vein cavernous transformation | Venous occlusion |

Document:
Author:


Template No.: Reference: CS\_WI\_BS005



Statistical Analysis Plan 

| Deep vein thrombosis | Portal vein embolism | Venous operation |
|---|---|---|
| Deep vein thrombosis postoperative | Portal vein occlusion | Venous recanalisation |
| Device embolisation | Portal vein thrombosis | Venous repair |
| Device occlusion | Portosplenomesenteric venous thrombosis | Venous stent insertion |
| Device related thrombosis | Post procedural myocardial infarction | Venous thrombosis |
| Diplegia | Post procedural pulmonary embolism | Venous thrombosis in pregnancy |
| Directional Doppler flow tests abnormal | Post procedural stroke | Venous thrombosis limb |
| Disseminated intravascular coagulation | Post thrombotic syndrome | Venous thrombosis neonatal |
| Disseminated intravascular coagulation in newborn | Postinfarction angina | Vertebral artery occlusion |
| Embolia cutis medicamentosa | Postoperative thrombosis | Vertebral artery thrombosis |
| Embolic cerebellar infarction | Postpartum thrombosis | Vessel puncture site occlusion |
| Embolic cerebral infarction | Postpartum venous thrombosis | Vessel puncture site thrombosis |
| Embolic pneumonia | Precerebral artery embolism | Visceral venous thrombosis |
| Embolic stroke | Precerebral artery occlusion | Visual acuity reduced transiently |
| Embolism | Precerebral artery thrombosis | Visual midline shift syndrome |
| Embolism arterial | Profundaplasty | |
| | Prosthetic cardiac valve thrombosis | |
| | Prosthetic vessel implantation | |
| | AESI Category: Hepatic function abnormal | |
| Acquired antithrombin III deficiency | Gastric variceal ligation | Hypothromboplastinaemia |
| Acquired factor IX deficiency | Gastric varices | Icterus index increased |
| Acquired factor V deficiency | Gastric varices haemorrhage | Immune-mediated cholangitis |
| Acquired factor VIII deficiency | Gastrooesophageal variceal haemorrhage prophylaxis | Immune-mediated hepatic disorder |
| Acquired factor XI deficiency | Graft versus host disease in liver | Immune-mediated hepatitis |
| Acquired hepatocerebral degeneration | Guanase increased | International normalised ratio abnormal |
| Acquired protein S deficiency | Haemangioma of liver | International normalised ratio increased |
| Acute graft versus host disease in liver | Haemorrhagic hepatic cyst | Intestinal varices |
| Acute hepatic failure | Hepaplastin abnormal | Intestinal varices haemorrhage |

Document:
Author:


Reference: CS\_WI\_BS005

Template No.:



## Statistical Analysis Plan 

| Acute on chronic liver failure | Hepaplastin decreased | Ischaemic hepatitis |
|---|---|---|
| Acute yellow liver atrophy | Hepatectomy | Jaundice |
| Alanine aminotransferase abnormal | Hepatic adenoma | Jaundice cholestatic |
| Alanine aminotransferase increased | Hepatic angiosarcoma | Jaundice hepatocellular |
| Allergic hepatitis | Hepatic artery flow decreased | Kayser-Fleischer ring |
| Alloimmune hepatitis | Hepatic atrophy | Liver carcinoma ruptured |
| Ammonia abnormal | Hepatic calcification | Liver dialysis |
| Ammonia increased | Hepatic cancer | Liver disorder |
| Anti factor X activity abnormal | Hepatic cancer metastatic | Liver function test abnormal |
| Anti factor X activity decreased | Hepatic cancer recurrent | Liver function test decreased |
| Anti factor X activity increased | Hepatic cancer stage I | Liver function test increased |
| Antithrombin III decreased | Hepatic cancer stage II | Liver induration |
| Ascites | Hepatic cancer stage III | Liver injury |
| Aspartate aminotransferase abnormal | Hepatic cancer stage IV | Liver operation |
| Aspartate aminotransferase increased | Hepatic cirrhosis | Liver palpable |
| AST/ALT ratio abnormal | Hepatic cyst | Liver scan abnormal |
| Asterixis | Hepatic cyst ruptured | Liver tenderness |
| Autoimmune hepatitis | Hepatic cytolysis | Liver transplant |
| Bacterascites | Hepatic encephalopathy | Lupoid hepatic cirrhosis |
| Benign hepatic neoplasm | Hepatic encephalopathy prophylaxis | Lupus hepatitis |
| Benign hepatobiliary neoplasm | Hepatic enzyme abnormal | Magnetic resonance imaging hepatobiliary abnormal |
| | | Magnetic resonance proton density fat fraction |
| Bile output abnormal | Hepatic enzyme decreased | measurement |
| Bile output decreased | Hepatic enzyme increased | Mitochondrial aspartate aminotransferase increased |
| Biliary ascites | Hepatic failure | Mixed hepatocellular cholangiocarcinoma |
| Biliary cirrhosis | Hepatic fibrosis | Mixed liver injury |
| Biliary fibrosis | Hepatic function abnormal | Molar ratio of total branched-chain amino acid to tyrosine |
| Bilirubin conjugated abnormal | Hepatic haemangioma rupture | Nodular regenerative hyperplasia |
| Bilirubin conjugated increased | Hepatic hamartoma | Nonalcoholic fatty liver disease |

Document:
Author:


Reference: CS\_WI\_BS005

Template No.:



## Statistical Analysis Plan 

| Bilirubin excretion disorder | Hepatic hydrothorax | Non-alcoholic steatohepatitis |
|---|---|---|
| Bilirubin urine present | Hepatic hypertrophy | Non-cirrhotic portal hypertension |
| Biopsy liver abnormal | Hepatic hypoperfusion | Ocular icterus |
| Blood bilirubin abnormal | Hepatic infiltration eosinophilic | Oedema due to hepatic disease |
| Blood bilirubin increased | Hepatic lesion | Oesophageal varices haemorrhage |
| Blood bilirubin unconjugated increased | Hepatic lipoma | Parenteral nutrition associated liver disease |
| Blood fibrinogen abnormal | Hepatic mass | Perihepatic discomfort |
| Blood fibrinogen decreased | Hepatic necrosis | Peripancreatic varices |
| Blood thrombin abnormal | Hepatic neoplasm | Portal fibrosis |
| Blood thrombin decreased | Hepatic neuroendocrine tumour | Portal hypertension |
| Blood thromboplastin abnormal | Hepatic pain | Portal hypertensive colopathy |
| Blood thromboplastin decreased | Hepatic sequestration | Portal hypertensive enteropathy |
| Bromosulphthalein test abnormal | Hepatic steato-fibrosis | Portal hypertensive gastropathy |
| Cardiohepatic syndrome | Hepatic steatosis | Portal vein cavernous transformation |
| Child-Pugh-Turcotte score abnormal | Hepatic vascular resistance increased | Portal vein dilatation |
| Child-Pugh-Turcotte score increased | Hepatic venous pressure gradient abnormal | Portopulmonary hypertension |
| Cholaemia | Hepatic venous pressure gradient increased | Primary biliary cholangitis |
| Cholangiosarcoma | Hepatitis | Protein C decreased |
| Cholestasis | Hepatitis acute | Protein S abnormal |
| Cholestatic liver injury | Hepatitis cholestatic | Protein S decreased |
| Cholestatic pruritus | Hepatitis chronic active | Prothrombin level abnormal |
| Chronic graft versus host disease in liver | Hepatitis chronic persistent | Prothrombin level decreased |
| Chronic hepatic failure | Hepatitis fulminant | Prothrombin time abnormal |
| Chronic hepatitis | Hepatitis toxic | Prothrombin time prolonged |
| Coagulation factor decreased | Hepatobiliary cancer | Prothrombin time ratio abnormal |
| Coagulation factor IX level abnormal | Hepatobiliary cancer in situ | Prothrombin time ratio increased |
| Coagulation factor IX level decreased | Hepatobiliary cyst | Radiation hepatitis |
| Coagulation factor V level abnormal | Hepatobiliary disease | Regenerative siderotic hepatic nodule |
| Coagulation factor V level decreased | Hepatobiliary neoplasm | Renal and liver transplant |

Document:


Template No.: Reference: CS\_WI\_BS005



Statistical Analysis Plan 

| Coagulation factor VII level abnormal | Hepatobiliary scan abnormal | Retrograde portal vein flow |
|---|---|---|
| Coagulation factor VII level decreased | Hepatoblastoma | Reye's syndrome |
| Coagulation factor X level abnormal | Hepatoblastoma recurrent | Reynold's syndrome |
| Coagulation factor X level decreased | Hepatocellular carcinoma | Splenic varices |
| Coma hepatic | Hepatocellular foamy cell syndrome | Splenic varices haemorrhage |
| Computerised tomogram liver abnormal | Hepatocellular injury | Spontaneous bacterial peritonitis |
| Congestive hepatopathy | Hepatomegaly | Steatohepatitis |
| Cryptogenic cirrhosis | Hepatopulmonary syndrome | Steatohepatitis |
| Diabetic hepatopathy | Hepatorenal failure | Subacute hepatic failure |
| Drug-induced liver injury | Hepatorenal syndrome | Sugiura procedure |
| Duodenal varices | Hepatosplenomegaly | Thrombin time abnormal |
| Flood syndrome | Hepatotoxicity | Thrombin time prolonged |
| Focal nodular hyperplasia | Hyperammonaemia | Total bile acids increased |
| Foetor hepaticus | Hyperbilirubinaemia | Transaminases abnormal |
| Galactose elimination capacity test abnormal | Hypercholia | Transaminases increased |
| Galactose elimination capacity test decreased | Hyperfibrinolysis | Ultrasound liver abnormal |
| Gallbladder varices | Hypertransaminasaemia | Urine bilirubin increased |
| Gamma-glutamyltransferase abnormal | Hypocoagulable state | Varices oesophageal |
| Gamma-glutamyltransferase increased | Hypofibrinogenaemia | Varicose veins of abdominal wall |
| Gastric variceal injection | Hypothrombinaemia | White nipple sign |
| | | X-ray hepatobiliary abnormal |
| | AESI Category: Left ventricular ejection fraction | n decreased |
| Acute left ventricular failure | Cardiohepatic syndrome | Hepatojugular reflux |
| Acute pulmonary oedema | Cardiopulmonary failure | Left ventricular failure |
| Acute right ventricular failure | Cardiorenal syndrome | Low cardiac output syndrome |
| Cardiac asthma | Chronic left ventricular failure | Neonatal cardiac failure |
| Cardiac failure | Chronic right ventricular failure | Obstructive shock |
| Cardiac failure acute | Congestive hepatopathy | Pulmonary oedema |

| Document: | |
|---------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |



Statistical Analysis Plan 

| Cardiac failure chronic | Cor pulmonale | Pulmonary oedema neonatal |
|---|---|---|
| Cardiac failure congestive | Cor pulmonale acute | Radiation associated cardiac failure |
| Cardiac failure high output | Cor pulmonale chronic | Right ventricular ejection fraction decreased |
| Cardiogenic shock | Ejection fraction decreased | Right ventricular failure |
| | | Ventricular failure |

# APPENDIX 6. CLINICAL LABORATORY PARAMETERS CTCAE CRITERIA

| PARAM (SI Unit) | Нуро | Hyper | ATOXGR | | | |
|---|---|---|---|---|---|---|
| | | | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
| | | | Increase in >0 - 2 | Increase in >2 - 4 | Increase in >4 gm/dL | |
| | | | gm/dL above ULN or | gm/dL above ULN or | above ULN or above | |
| | | | above baseline if | above baseline if | baseline if baseline is | |
| | | Hemoglobin | baseline is above ULN | baseline is above | above ULN | |
| | | increased | | ULN | · | ~ |
| | | | Hemoglobin (Hgb) | | | |
| | | | <lln -="" 10.0="" dl;<="" g="" td=""><td>Hgb &lt; 10.0 - 8.0 g/dL;</td><td></td><td></td></lln> | Hgb < 10.0 - 8.0 g/dL; | | |
| | | | <lln -="" 6.2="" l;<="" mmol="" td=""><td>&lt;6.2 - 4.9 mmol/L;</td><td>Hgb &lt;8.0 g/dL; &lt;4.9</td><td></td></lln> | <6.2 - 4.9 mmol/L; | Hgb <8.0 g/dL; <4.9 | |
| Hemoglobin (g/L) | Anemia | | <lln -="" 100="" g="" l<="" td=""><td>&lt;100 - 80g/L</td><td>mmol/L; &lt;80 g/L</td><td>~</td></lln> | <100 - 80g/L | mmol/L; <80 g/L | ~ |
| | | | | <75,000 - | <50,000 - | |
| | Platelet count | | <lln -="" 75,000="" mm3;<="" td=""><td>50,000/mm3; &lt;75.0 -</td><td>25,000/mm3; &lt;50.0 -</td><td>&lt;25,000/mm3;</td></lln> | 50,000/mm3; <75.0 - | 25,000/mm3; <50.0 - | <25,000/mm3; |
| Platelets (10 <sup>9</sup> /L) | decreased | | <lln -="" 10e9="" 75.0="" l<="" td="" x=""><td>50.0 x 10e9 /L</td><td>25.0 x 10e9 /L</td><td>&lt;25.0 x 10e9 /L</td></lln> | 50.0 x 10e9 /L | 25.0 x 10e9 /L | <25.0 x 10e9 /L |
| | | | | | | 1000/ |
| | White blood cell | | <lln -="" 3000="" mm3;<="" td=""><td>&lt;3000 - 2000/mm3;</td><td>&lt;2000 - 1000/mm3;</td><td>&lt;1000/mm3;</td></lln> | <3000 - 2000/mm3; | <2000 - 1000/mm3; | <1000/mm3; |
| Leukocytes (10^9/L) | decreased | | <lln -="" 10e9="" 3.0="" l<="" td="" x=""><td>&lt;3.0 - 2.0 x 10e9 /L</td><td>&lt;2.0 - 1.0 x 10e9 /L</td><td>&lt;1.0 x 10e9 /L</td></lln> | <3.0 - 2.0 x 10e9 /L | <2.0 - 1.0 x 10e9 /L | <1.0 x 10e9 /L |

| Document: | |
|---------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |

Effective Date: 02Dec2019

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



Statistical Analysis Plan 

| Neutrophils (10^9/L) | Neutrophil count decreased | | <lln -="" 1500="" mm3;<br=""><lln -="" 1.5="" 10e9="" l<="" th="" x=""><th>&lt;1500 - 1000/mm3;<br/>&lt;1.5 - 1.0 x 10e9 /L</th><th>&lt;1000 - 500/mm3;<br/>&lt;1.0 - 0.5 x 10e9 /L</th><th>&lt;500/mm3; &lt;0.5<br/>x 10e9 /L</th></lln></lln> | <1500 - 1000/mm3;<br><1.5 - 1.0 x 10e9 /L | <1000 - 500/mm3;<br><1.0 - 0.5 x 10e9 /L | <500/mm3; <0.5<br>x 10e9 /L |
|---|---|---|---|---|---|---|
| | Lymphocyte count decreased | | <lln -="" 800="" mm3;<br=""><lln -="" 0.8="" 10e9="" l<="" td="" x=""><td>&lt;800 - 500/mm3;<br/>&lt;0.8 - 0.5 x 10e9 /L</td><td>&lt;500 - 200/mm3;<br/>&lt;0.5 - 0.2 x 10e9 /L</td><td>&lt;200/mm3; &lt;0.2<br/>x 10e9 /L</td></lln></lln> | <800 - 500/mm3;<br><0.8 - 0.5 x 10e9 /L | <500 - 200/mm3;<br><0.5 - 0.2 x 10e9 /L | <200/mm3; <0.2<br>x 10e9 /L |
| Lymphocytes (10^9/L) | | Lymphocyte count increased | ~ | >4000/mm3 -<br>20,000/mm3 | >20,000/mm3 | ~ |
| Activated Partial<br>Thromboplastin Time (s) | | Activated partial thromboplastin time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; bleeding | ~ |
| International Normalized Ratio | | INR increased | >1.2 - 1.5 | >1.5 - 2.5 | >2.5 | ~ |
| Albumin (g/L) | Hypoalbuminemia | | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>~</td></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | ~ |
| Glucose (mmol/L) | Hypoglycemia | | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 - 40 mg/dL; &lt;3.0 - 2.2 mmol/L</td><td>&lt;40 - 30 mg/dL; &lt;2.2<br/>- 1.7 mmol/L</td><td>&lt;30 mg/dL; &lt;1.7 mmol/L</td></lln></lln> | <55 - 40 mg/dL; <3.0 - 2.2 mmol/L | <40 - 30 mg/dL; <2.2<br>- 1.7 mmol/L | <30 mg/dL; <1.7 mmol/L |
| Creatinine (umol/L) | | Creatinine increased | >1 - 1.5 x<br>baseline; >ULN - 1.5 x<br>ULN | >1.5 - 3.0 x<br>baseline; >1.5 - 3.0 x<br>ULN | >3.0 baseline; >3.0 -<br>6.0 x ULN | >6.0 x ULN |
| Alkaline Phosphatase (IU/L) | | Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |

| Document: | |
|---------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |



Statistical Analysis Plan 

| Aspartate Aminotransferase (IU/L) | | Aspartate<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
|---|---|---|---|---|---|---|
| Alanine Aminotransferase (IU/L) | | Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| | | Hypercalcemia | >ULN - 2.9 mmol/L | >2.9 - 3.1 mmol/L | >3.1 - 3.4 mmol/L | >3.4 mmol/L |
| Serum Calcium (mmol/L) | Hypocalcemia | | <lln -="" 2.0="" l<="" mmol="" td=""><td>&lt;2.0 - 1.75 mmol/L</td><td>&lt;1.75 - 1.5 mmol/L</td><td>&lt;1.5 mmol/L</td></lln> | <2.0 - 1.75 mmol/L | <1.75 - 1.5 mmol/L | <1.5 mmol/L |
| | | Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | ~ | >3.0 - 8.0 mg/dL;<br>>1.23 - 3.30 mmol/L | >8.0 mg/dL;<br>>3.30 mmol/L |
| Magnesium (mmol/L) | Hypomagnesemia | | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 - 0.7 mg/dL;<br/>&lt;0.4 - 0.3 mmol/L</td><td>&lt;0.7 mg/dL; &lt;0.3 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL;<br><0.4 - 0.3 mmol/L | <0.7 mg/dL; <0.3 mmol/L |
| | | Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L | >7.0 mmol/L |
| Potassium (mmol/L) | Hypokalemia | | <lln -="" 3.0="" l<="" mmol="" td=""><td>~</td><td>&lt;3.0 - 2.5 mmol/L</td><td>&lt;2.5 mmol/L</td></lln> | ~ | <3.0 - 2.5 mmol/L | <2.5 mmol/L |
| | | Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L | >160 mmol/L |
| Sodium (mmol/L) | Hyponatremia | | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L</td></lln> | - | <130 - 120 mmol/L | <120 mmol/L |
| Total cholesterol (mmol/L) | | Cholesterol high | >ULN - 300 mg/dL;<br>>ULN - 7.75 mmol/L | >300 - 400 mg/dL;<br>>7.75 - 10.34 mmol/L | >400 - 500 mg/dL;<br>>10.34 - 12.92<br>mmol/L | >500 mg/dL;<br>>12.92 mmol/L |

| Document: | |
|---------------|------------------------|
| Template No.: | Reference: CS_WI_BS005 |



Statistical Analysis Plan 

| Bilirubin (umol/L) | Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN |
|---|---|---|---|---|---|
| Triglycerides (mmol/L) | | 150 mg/dL - 300<br>mg/dL; 1.71 mmol/L -<br>3.42 mmol/L | >300 mg/dL - 500<br>mg/dL; >3.42 mmol/L<br>- 5.7 mmol/L | >500 mg/dL - 1000<br>mg/dL; >5.7 mmol/L<br>- 11.4 mmol/L | >1000 mg/dL;<br>>11.4 mmol/L |
| Urinary protein | Proteinuria | 1+ proteinuria; urinary<br>protein <1.0 g/24 hrs | 2+ proteinura; urinary<br>protein 1.0 -<br>3.4g/24hrs | urinary protein >= 3.5g/24hrs | ~ |

Document:
Author:


Template No.: Reference: CS\_WI\_BS005